CLINICAL TRIAL: NCT03191864
Title: FLUTicasone in Eosinophilic Esophagitis (FLUTE): A Randomized, Double-blind, Placebo-controlled, Dose-ranging, and Maintenance Study of APT-1011 in Subjects With Eosinophilic Esophagitis
Brief Title: Efficacy, Safety, and Pharmacokinetics of APT-1011 in Subjects With Eosinophilic Esophagitis (EoE)
Acronym: FLUTE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Adare Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP-1011-002; 2016-004749-10 (EudraCT Number)
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Results first posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Eosinophilic Esophagitis
Keywords: Esophagitis; Eosinophilic Esophagitis; Fluticasone; Dysphagia; Safety; Efficacy; Pharmacokinetics; Esophageal Diseases; Gastrointestinal Diseases; Digestive System Diseases; Glucocorticoids; Orally Disintegrating Tablet
MeSH Terms: conditions — Eosinophilic Esophagitis; Esophagitis; Deglutition Disorders; Esophageal Diseases; Gastrointestinal Diseases; Digestive System Diseases | interventions — APT-1011

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- APT-1011 1.5 mg HS (Experimental): Placebo after breakfast, APT-1011 1.5 mg HS
  Interventions: Drug: APT-1011; Drug: Placebo
- APT-1011 1.5 mg BID (Experimental): APT-1011 1.5 mg after breakfast, APT-1011 1.5 mg HS
  Interventions: Drug: APT-1011
- APT-1011 3 mg HS (Experimental): Placebo after breakfast, APT-1011 3 mg HS
  Interventions: Drug: APT-1011; Drug: Placebo
- APT-1011 3 mg BID (Experimental): APT-1011 3 mg after breakfast, APT-1011 3 mg HS
  Interventions: Drug: APT-1011
- Placebo BID (Placebo Comparator): Placebo 30 minutes after breakfast and HS
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APT-1011 — APT-1011 is an orally disintegrating tablet formulation of fluticasone propionate
  Other Names: Fluticasone propionate ODT
  Arms: APT-1011 1.5 mg BID; APT-1011 1.5 mg HS; APT-1011 3 mg BID; APT-1011 3 mg HS
Drug: Placebo — Placebo tablets are identical in composition to APT-1011 except they exclude the active ingredient.
  Other Names: Matching placebo dose
  Arms: APT-1011 1.5 mg HS; APT-1011 3 mg HS; Placebo BID

SUMMARY:
Eosinophilic esophagitis (EoE) is an inflammatory disease of the esophagus, characterized by eosinophilic infiltration and gastrointestinal symptoms. Swallowed, topically acting corticosteroids, such as fluticasone, appear to be effective in resolving acute clinical and pathological features of EoE.

APT-1011 is an orally disintegrating tablet (ODT) formulation of fluticasone propionate. This study is designed to compare the efficacy and safety of APT-1011 with placebo in adults with EoE for an initial 12-week treatment period, followed by an additional 40-week maintenance treatment phase. Histologic response, pharmacokinetics, and dysphagia will be assessed.

DETAILED DESCRIPTION:
FLUTE is a phase 2b randomized, double-blind, placebo-controlled dose-ranging clinical trial of APT-1011 versus placebo in 100 adult subjects (≥18 years of age) diagnosed with EoE. Efficacy (including histologic, endoscopic, and symptomatic response), safety, and PK of APT-1011 will be examined. Participants will be given an electronic diary to record symptoms and medication intake daily.

FLUTE will be conducted in several parts (Screening [4 weeks], followed by a 4-week Baseline Symptom Assessment, and 2 treatment parts [Part 1: 14-week Induction and Part 2: 38-week Maintenance]), with a follow-up visit to occur 2 weeks after the final dose of study drug.

In Part 1 of the study, approximately 100 subjects will be randomized 1:1:1:1:1 to receive placebo or one of 4 active doses of APT-1011. All subjects will receive one tablet 30 minutes after breakfast and one tablet at bedtime (HS). The dosing groups include: 1.5 mg HS APT-1011, 1.5 mg twice daily (BID) (total daily dose of 3 mg) APT-1011, 3 mg HS APT-1011, and 3 mg BID (total daily dose of 6 mg) APT-1011, and placebo BID.

In Part 2, all subjects classified as histologic responders at Week 12 will continue to be treated according to the dosing group to which they were randomized, and non-responders will receive single-blind 3 mg BID. All subjects who are histologic non-responders at Week 26 will stop treatment at Week 28 and enter the 2-week follow-up and exit the study. Histologic responders at Week 26 will continue on the same dose until end-of-study at Week 52.

Subjects will complete a follow-up visit 2 weeks after the final dose of study drug. All subjects must have a final EGD within 3 weeks prior to completing the Follow-up Visit unless the subject withdraws consent or has a contraindication to EGD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between ≥18 and ≤75 years of age at the time of informed consent
* Signed informed consent
* Evidence of EoE defined by ≥15 peak eosinophils per HPF as measured from proximal and distal biopsies
* Subject-reported history of ≥3 episodes of dysphagia in the 7 days prior to Screening
* 7-day Global EoE Symptom Score >3 at baseline and at screening
* Willing and able to adhere to study-related treatment regimens, procedures, and visit schedule

Exclusion Criteria:

* Have known contraindication, hypersensitivity, or intolerance to corticosteroids;
* Have any physical, mental, or social condition or history of illness or laboratory abnormality that in the Investigator's judgment might interfere with study procedures or the ability of the subject to adhere to and complete the study;
* Presence of oral or esophageal mucosal infection of any type;
* Have any mouth or dental condition that prevents normal eating;
* Have any condition affecting the esophageal mucosa or altering esophageal motility other than EoE;
* Use of systemic corticosteroids within 60 days prior to Screening, use of inhaled/swallowed corticosteroids within 30 days prior to Screening, or extended use of high-potency dermal topical corticosteroids within 30 days prior to Screening;
* Initiation of an elimination diet or elemental diet within 30 days before Screening (diet must remain stable after signing ICF);
* Morning serum cortisol level ≤5 μg/dL (138 nmol/L);
* Use of biologic immunomodulators in the 24 weeks prior to Screening;
* Use of calcineurin inhibitors or purine analogues, or potent cytochrome P450 (CYP) 3A4 inhibitors in the 12 weeks prior to Screening;
* Have a contraindication to or factors that substantially increase the risk of EGD or esophageal biopsy or have narrowing of the esophagus that precludes EGD with a standard 9 mm endoscope;
* Have a history of an esophageal stricture requiring dilatation within the previous 12 weeks prior to Screening;
* Have initiated, discontinued or changed dosage regimen of PPIs, H2 antagonists, antacids or antihistamines for any condition such as GERD or allergic rhinitis within 4 weeks prior to qualifying endoscopy. These drugs must remain constant throughout the study.
* A serum cortisol level <18 μg/dL (497 nmol/L) at 60 minutes with adrenocorticotropic hormone (ACTH) stimulation test using 250 μg cosyntropin (i.e., a positive result on the ACTH stimulation test).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Richardson, Study Director — Adare Pharmaceuticals, Inc.
Locations (75):
- United States (51):
  - Del Sol Research Management, LLC, Chandler, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Arkansas Gastroenterology, P.A., Sherwood, Arkansas
  - Hope Clinical Research, Canoga Park, California
  - TriWest Research Associates, LLC, El Cajon, California
  - SC Clinical Research, Inc., Garden Grove, California
  - Beverly Hills Center for Digestive Health, Los Angeles, California
  - Focilmed, Oxnard, California
  - Precision Research Institute, LLC, San Diego, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Care Access Research LLC, San Pablo, California
  - Stanford University School of Medicine, Stanford, California
  - St. Jude Healthcare, Yorba Linda, California
  - Western Connecticut Health Network, Danbury, Connecticut
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Eastern Research, Inc., Hialeah, Florida
  - Nature Coast Clinical Research, LLC, Inverness, Florida
  - Sunrise Medical Research, Lauderdale Lakes, Florida
  - DBC Research, Corp, Pembroke Pines, Florida
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - Rockford Gastroenterology Associates, Ltd., Rockford, Illinois
  - MediSphere Medical Research Center, an AMR affiliate, Evansville, Indiana
  - Cotton-O'Neil Clinical Research Center, Digestive Health, Topeka, Kansas
  - Gastroenterology Associates, Hazard, Kentucky
  - Clinical Trials of America, Inc., West Monroe, Louisiana
  - Henry Ford Medical Center, Novi, Michigan
  - Metro Health, Wyoming, Michigan
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - Long Island Gastrointestinal Research Group, LLP, Great Neck, New York
  - Weill Cornell Medical College, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Research Institute of the Carolinas, PLC, Mooresville, North Carolina
  - Carolina's GI Research, LLC, Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - PMG Research of Salisbury, LLC, Salisbury, North Carolina
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Aventiv Research Inc., Columbus, Ohio
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - Allergy and Asthma Center of South Oregon, Medford, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Digestive Disease Associates, Ltd., Wyomissing, Pennsylvania
  - Rapid City Medical Center, LLP, Rapid City, South Dakota
  - Advanced Gastroenterology, Union City, Tennessee
  - Avant Research Associates, LLC - Austin, Austin, Texas
  - Avant Research Associates, LLC, Beaumont, Texas
  - DHAT Research Institute, Richardson, Texas
  - Advanced Research Institute, Ogden, Utah
  - University of Utah, Salt Lake City, Utah
  - Care Access Research LLC, Salt Lake City, Utah
  - Verity Research Inc, Fairfax, Virginia
- Belgium (4):
  - AZ Sint-Lucas, Bruges
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Groeninge - Kennedylaan, Kortrijk
  - UZ Leuven, Leuven
- Canada (5):
  - (G.I.R.I.) GI Research Institute, Vancouver, British Columbia
  - Viable Clinical Research, Bridgewater, Nova Scotia
  - Viable Clinical Research, Lindsay, Ontario
  - London Health Science Centre, London, Ontario
  - Taunton Surgical Centre, Oshawa, Ontario
- Germany (5):
  - Klinikum rechts der Isar der TU Muenchen, Munich, Bavaria
  - Staedisches Klinikum Brandenburg, Brandenburg, Brandenburg
  - Praxis am Germania, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Leipzig AoeR, Leipzig, Saxony
  - Universitaetsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
- Spain (9):
  - Hospital General de Tomelloso, Tomelloso, Ciudad Real
  - Hospital General Universitario de Alicante, Alicante
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dellon ES, Lucendo AJ, Schlag C, Schoepfer AM, Falk GW, Eagle G, Nezamis J, Comer GM, Knoop K, Hirano I. Fluticasone Propionate Orally Disintegrating Tablet (APT-1011) for Eosinophilic Esophagitis: Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2022 Nov;20(11):2485-2494.e15. doi: 10.1016/j.cgh.2022.02.013. Epub 2022 Feb 16. PMID 35181572

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment in 6 countries (United States, Canada, Belgium, Germany, Spain, and Switzerland) took place between 22-Jun-2017 (First Subject Enrolled) until 23-Aug-2018 (Last Subject Enrolled).
Pre-assignment Details: The Screening Period was 4 weeks (28 days) and utilized a single-blind placebo run-in period. Along with the reports confirming the subject's primary diagnosis of EoE, the Investigator assessed eligibility criteria of the subject based on screening results. The Global EoE Symptom Score had to be >3 for the subject to continue in the study.
  Patients who were screened (308) are presented under Baseline Symptom Assessment, those enrolled (106) are presented in Part 1 - Induction.
Groups:
- Single-blind APT-1011 3mg BID: APT-1011 3 mg after breakfast, APT-1011 3 mg HS
  APT-1011: APT-1011 is an orally disintegrating tablet formulation of fluticasone propionate
Period: Baseline Symptom Assessment
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Single-blind APT-1011 3mg BID | Placebo BID
Started (Due to the high placebo response rates, the study utilized a 4-week single-blind placebo run-in period to not only establish the baseline symptoms for the study, but also to ensure that all subjects enrolled had sufficient severity of EoE to warrant inclusion in the study.) | 0 | 0 | 0 | 0 | 0 | 308
Completed | 0 | 0 | 0 | 0 | 0 | 106
Not Completed | 0 | 0 | 0 | 0 | 0 | 202
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Patient Diary Unavailable at Site | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 19
Not completed — Violation of inclusion/exclusion criteria | 0 | 0 | 0 | 0 | 0 | 179
Period: Part 1 - Induction
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Single-blind APT-1011 3mg BID | Placebo BID
Started | 21 | 22 | 22 | 20 | 0 | 21
Completed | 18 | 19 | 20 | 19 | 0 | 16
Not Completed | 3 | 3 | 2 | 1 | 0 | 5
Not completed — Violation of inclusion/exclusion criteria | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 2 | 0 | 1 | 0 | 2
Not completed — Randomized but never dosed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 0 | 0 | 2
Period: Part 2 - Maintenance
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Single-blind APT-1011 3mg BID | Placebo BID
Started (Note that those subjects that were non-responders at Week 12 were switched from another arm to the Single-blind APT-1011 3 mg BID arm. This arm was a single-blinded arm for the subjects only.) | 10 | 19 | 14 | 16 | 34 | 0
Completed | 5 | 17 | 11 | 14 | 19 | 0
Not Completed | 5 | 2 | 3 | 2 | 15 | 0
Not completed — Refused EGD at Week 26 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Subject Could Not Transfer Site to Complete the Study | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 2 | 2 | 2 | 10 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 3 | 0
Not completed — Unresponsive - Patient missed multiple appointments | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Placebo BID | Total
Number analyzed (Participants) | 21 | 22 | 22 | 20 | 21 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 21 | 20 | 21 | 104
  >=65 years | 0 | 1 | 1 | 0 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (11.65) | 41.3 (12.24) | 41.9 (12.09) | 36.8 (9.19) | 38.7 (13.94) | 39.2 (11.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 10 | 4 | 5 | 33
  Male | 14 | 15 | 12 | 16 | 16 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 2 | 2 | 3 | 16
  Not Hispanic or Latino | 17 | 17 | 20 | 16 | 17 | 87
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 1 | 3
  White | 21 | 22 | 21 | 19 | 20 | 103
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  North America | 15 | 16 | 18 | 13 | 17 | 79
  Europe | 6 | 6 | 4 | 7 | 4 | 27
Smoking Status [Count of Participants; unit: Participants]
  Never | 18 | 17 | 19 | 16 | 17 | 87
  Former | 2 | 3 | 3 | 4 | 4 | 16
  Current | 1 | 2 | 0 | 0 | 0 | 3
  Missing | 0 | 0 | 0 | 0 | 0 | 0
History of esophageal stricture(s) [Count of Participants; unit: Participants]
  Yes | 11 | 10 | 8 | 8 | 9 | 46
  No | 10 | 12 | 14 | 12 | 12 | 60
  Missing | 0 | 0 | 0 | 0 | 0 | 0
Current esophageal stricture(s) based on the study EGD [Count of Participants; unit: Participants]
  Yes | 4 | 5 | 5 | 4 | 5 | 23
  No | 17 | 17 | 17 | 16 | 16 | 83
  Missing | 0 | 0 | 0 | 0 | 0 | 0
History of positive steroid response to EOE [Count of Participants; unit: Participants]
  Yes | 3 | 5 | 5 | 4 | 4 | 21
  No | 18 | 17 | 17 | 16 | 17 | 85
  Missing | 0 | 0 | 0 | 0 | 0 | 0
Proton pump inhibitor status [Count of Participants; unit: Participants]
  Continuing into study | 12 | 16 | 13 | 11 | 14 | 66
  Not continuing into study | 9 | 6 | 9 | 9 | 7 | 40
  Missing | 0 | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 175.4 (8.55) | 173.0 (8.56) | 171.0 (9.62) | 176.7 (8.61) | 174.8 (7.20) | 174.1 (8.63)
Weight [Mean (Standard Deviation); unit: kg] | 87.45 (17.69) | 83.72 (14.72) | 83.47 (18.45) | 79.72 (14.93) | 85.45 (19.79) | 83.96 (17.09)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.27 (5.19) | 27.39 (4.34) | 28.68 (6.74) | 25.54 (4.45) | 28.02 (6.53) | 27.60 (5.57)
Global EOE Symptom Score prior to randomization [Mean (Standard Deviation); unit: units on a scale] — Global Eosinophilic Esophagitis Symptom Score: On a scale from 0 (no symptoms) to 10 (most severe symptoms), how severe were your EoE symptoms over the past 7 days? Patients were asked to think of all their symptoms due to EoE and make an overall statement by selecting a number.
  units on a scale | 5.14 (1.62) | 4.50 (2.13) | 5.00 (1.95) | 4.25 (1.94) | 4.95 (1.66) | 4.77 (1.87)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With ≤6 Peak Eosinophils/High-power Field (HPF)
Description: Histology (eosinophils per high power field [HPF]): percentage of subjects with ≤6 PEAK eosinophils/HPF after assessing at least 5-6 biopsies from the proximal and distal esophagus (~3 each) where the HPF area is 235 square microns (40 magnification lens with a 22 mm ocular).
Time Frame: Week 12
Population: Full Analysis Set Population
Measure: Count of Participants; unit: Participants
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Placebo BID
Number analyzed (Participants) | 21 | 22 | 21 | 20 | 19
Participants
  Responder | 10 | 19 | 14 | 16 | 0
  Non-Responder | 11 | 3 | 7 | 4 | 19
Statistical Analysis 1: Comparison: APT-1011 1.5 mg HS vs Placebo BID; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: APT-1011 1.5 mg BID vs Placebo BID; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: APT-1011 3 mg HS vs Placebo BID; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: APT-1011 3 mg BID vs Placebo BID; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Percentage of Subjects Who Met the Primary Endpoint at Week 12 and Maintained the Primary Endpoint at Weeks 26 and 52
Description: Percentage of subjects who entered Part 2 - Maintenance and met the primary endpoint (histology) at Week 12 and maintained the primary endpoint at Week 26 and Week 52.
  Note: Following Week 14, all patients in the placebo group were given APT-1011 3mg BID and results reflect percentage of subjects who met the primary endpoint following 12 or 38 weeks of treatment.
Time Frame: Week 26, and Week 52
Population: Full Analysis Set Population
Measure: Count of Participants; unit: Participants
Groups:
- Responder APT-1011 1.5 mg HS: Placebo after breakfast, APT-1011 1.5 mg HS
  APT-1011: APT-1011 is an orally disintegrating tablet formulation of fluticasone propionate
  Placebo: Placebo tablets are identical in composition to APT-1011 except they exclude the active ingredient.
- Responder APT-1011 1.5 mg BID: APT-1011 1.5 mg after breakfast, APT-1011 1.5 mg HS
  APT-1011: APT-1011 is an orally disintegrating tablet formulation of fluticasone propionate
- Responder APT-1011 3 mg HS: Placebo after breakfast, APT-1011 3 mg HS
  APT-1011: APT-1011 is an orally disintegrating tablet formulation of fluticasone propionate
  Placebo: Placebo tablets are identical in composition to APT-1011 except they exclude the active ingredient.
- Responder APT-1011 3 mg BID: APT-1011 3 mg after breakfast, APT-1011 3 mg HS
  APT-1011: APT-1011 is an orally disintegrating tablet formulation of fluticasone propionate
- Non-Responder APT-1011, APT-1011 3mg BID (Part 2): APT-1011 3 mg after breakfast, APT-1011 3 mg HS
  All Non-responders at Week 12 received 3 mg BID Week 14 to Week 52
- Placebo BID, APT-1011 3 mg BID (Part 2): Placebo 30 minutes after breakfast and HS
  All Non-responders at Week 12 received 3 mg BID Week 14 to Week 52
Arm/Group | Responder APT-1011 1.5 mg HS | Responder APT-1011 1.5 mg BID | Responder APT-1011 3 mg HS | Responder APT-1011 3 mg BID | Non-Responder APT-1011, APT-1011 3mg BID (Part 2) | Placebo BID, APT-1011 3 mg BID (Part 2)
Number analyzed (Participants) | 10 | 19 | 14 | 16 | 18 | 16
Participants
  Week 26 Responders | 7 | 17 | 11 | 14 | 7 | 12
  Week 52 Responders | 3 | 16 | 9 | 11 | 5 | 10

3. Secondary Outcome: Change From Baseline Eosinophilic Esophagitis Endoscopic Reference Score (EREFs) at Week 12, 26, and 52
Description: Endoscopic changes will be assessed as per the EREFs evaluation based on the following endoscopic features: edema [Grade {Gr} 0 (absent) or Gr 1 (present)], strictures [Gr 0 (absent) or Gr 1 (present)], rings [Gr 0 (none), Gr 1 (mild), Gr 2 (moderate), Gr 3 (severe)], exudates [Gr 0 (none), Gr 1 (mild), Gr (severe)], furrows [Gr 0 (none), Gr 1 (mild), Gr 2 (severe)], crepe paper esophagus [Gr 0 (absent) or Gr 1 (present)], narrow caliber esophagus [Gr 0 (absent) or Gr 1 (present)], and esophageal erosions [Normal (0), Gr A (1), Gr B (2), Gr C (3), or Gr D (4)].
  EREFs: 0 (best) to 15 (worst) based on the sum of the subscores listed above.
  Population used are those who entered Part 1 - Induction. The number of participants analyzed for each timepoint reflect the actual number of participants with data at that timepoint. Note: Following Week 14, all patients in the placebo group were given APT-1011 3 mg BID and results reflect EREF evaluation following 12 or 38 weeks of treatment.
Time Frame: Week 12, Week 26, and Week 52
Population: Full Analysis Set Population receiving double-blind study medication
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Placebo BID
Number analyzed (Participants) | 18 | 20 | 20 | 19 | 17
units on a scale
  Week 12 Change From Baseline | -2.4 (2.04) | -2.7 (2.66) | -3.3 (2.36) | -2.2 (2.15) | -0.9 (1.62)
  Week 26 Change From Baseline: number analyzed (Participants) | 8 | 19 | 13 | 16 | 0
  Week 26 Change From Baseline | -3.1 (1.25) | -3.2 (2.77) | -4.2 (2.61) | -3.0 (1.67) |
  Week 52 Change From Baseline: number analyzed (Participants) | 5 | 17 | 11 | 14 | 0
  Week 52 Change From Baseline | -3.4 (1.82) | -3.5 (3.08) | -3.8 (3.19) | -2.9 (1.29) |
Statistical Analysis 1: Comparison: APT-1011 1.5 mg HS vs Placebo BID; Least-squares Mean differences, 90% confidence intervals and 1-sided p-values for comparisons of each APT-1011 dose group to Placebo at Week 12 are from an ANCOVA model; Test type: Other; p = 0.020, ANCOVA; Mean Difference (Final Values) = -1.28, 90% CI 2-sided [-2.29 to -0.26]
Statistical Analysis 2: Comparison: APT-1011 1.5 mg BID vs Placebo BID; [analysis description as in outcome 3, analysis 1]; Test type: Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -2.08, 90% CI 2-sided [-3.07 to -1.10]
Statistical Analysis 3: Comparison: APT-1011 3 mg HS vs Placebo BID; [analysis description as in outcome 3, analysis 1]; Test type: Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -2.25, 90% CI 2-sided [-3.23 to -1.26]
Statistical Analysis 4: Comparison: APT-1011 3 mg BID vs Placebo BID; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.005, ANCOVA; Mean Difference (Final Values) = -1.59, 90% CI 2-sided [-2.59 to -0.59]

4. Secondary Outcome: Percentage of Subjects With a Peak Eosinophils/HPF Number <1 and <15
Description: Percentage of subjects with a peak eosinophils/HPF <1 and <15 at Week 12, 26 and 52.
  Population used are those who entered Part 1 - Induction. The number of participants analyzed for each timepoint reflect the actual number of participants with data at that timepoint. Note: Following Week 14, all patients in the placebo group were given APT-1011 3mg BID and results reflect peak eosinophils/HPF following 12 or 38 weeks of treatment.
Time Frame: Week 12, Week 26, and Week 52
Population: Full Analysis Set Population receiving double-blind study medication
Measure: Count of Participants; unit: Participants
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Placebo BID
Number analyzed (Participants) | 18 | 20 | 20 | 19 | 17
Participants
  Week 12 : <1/HPF | 7 | 14 | 12 | 15 | 0
  Week 12 : <15/HPF | 12 | 19 | 15 | 16 | 1
  Week 26 : <1/HPF: number analyzed (Participants) | 8 | 19 | 13 | 16 | 0
  Week 26 : <1/HPF | 4 | 15 | 9 | 13 |
  Week 26 : <15/HPF: number analyzed (Participants) | 8 | 19 | 13 | 19 | 0
  Week 26 : <15/HPF | 8 | 18 | 12 | 14 |
  Week 52 : <1/HPF: number analyzed (Participants) | 5 | 17 | 11 | 14 | 0
  Week 52 : <1/HPF | 1 | 12 | 7 | 10 |
  Week 52 : <15/HPF: number analyzed (Participants) | 5 | 17 | 11 | 14 | 0
  Week 52 : <15/HPF | 3 | 17 | 10 | 12 |

5. Secondary Outcome: Change From Baseline Global EoE Symptom Score
Description: Change from baseline global EOE symptom score assessed prior to randomization to scores for 7-day recall at Week 4, 8, 12, 14, 18, 22, 26, 28, 36, 44, and 52 visits.
  Global Eosinophilic Esophagitis Symptom Score: On a scale from 0 (no symptoms) to 10 (most severe symptoms), how severe were your EoE symptoms over the past 7 days? Patients were asked to think of all their symptoms due to EoE and make an overall statement by selecting a number.
  Population used are those who entered Part 1 - Induction. The number of participants analyzed for each timepoint reflect the actual number of participants with data at that timepoint. Note: Following Week 14, all patients in the placebo group were given APT-1011 3mg BID and results reflect change from baseline global EOE symptom score following 4, 8, 12, 14, 22, 30 or 38 weeks of treatment.
Time Frame: Week 4, 8, 12, 14, 18, 22, 26, 28, 36, 44, and 52
Population: Full Analysis Set Population receiving double-blind study medication
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Placebo BID
Number analyzed (Participants) | 21 | 21 | 20 | 20 | 17
units on a scale
  Week 4 Change from Baseline: number analyzed (Participants) | 21 | 20 | 20 | 20 | 16
  Week 4 Change from Baseline | -1.8 (2.64) | -1.3 (2.15) | -2.5 (3.12) | -1.6 (1.39) | -1.0 (1.67)
  Week 8 Change from Baseline: number analyzed (Participants) | 18 | 21 | 19 | 20 | 17
  Week 8 Change from Baseline | -2.6 (2.12) | -1.7 (1.94) | -3.1 (2.64) | -2.1 (1.92) | -1.4 (2.21)
  Week 12 Change from Baseline: number analyzed (Participants) | 18 | 21 | 20 | 19 | 17
  Week 12 Change from Baseline | -3.1 (2.17) | -1.5 (2.20) | -3.1 (2.74) | -1.7 (2.42) | -1.7 (1.83)
  Week 14 Change from Baseline: number analyzed (Participants) | 10 | 18 | 13 | 16 | 0
  Week 14 Change from Baseline | -2.7 (2.26) | -2.3 (2.45) | -3.9 (2.81) | -2.8 (1.77) |
  Week 18 Change from Baseline: number analyzed (Participants) | 9 | 19 | 14 | 15 | 0
  Week 18 Change from Baseline | -4.1 (1.36) | -2.7 (2.58) | -4.1 (2.92) | -3.1 (2.17) |
  Week 22 Change from Baseline: number analyzed (Participants) | 8 | 19 | 14 | 16 | 0
  Week 22 Change from Baseline | -4.0 (1.41) | -3.2 (2.46) | -3.8 (2.97) | -3.0 (2.76) |
  Week 26 Change from Baseline: number analyzed (Participants) | 8 | 18 | 13 | 16 | 0
  Week 26 Change from Baseline | -3.8 (1.39) | -3.1 (2.52) | -4.0 (2.68) | -3.8 (2.57) |
  Week 28 Change from Baseline: number analyzed (Participants) | 7 | 18 | 10 | 14 | 0
  Week 28 Change from Baseline | -4.3 (1.38) | -3.3 (2.42) | -4.8 (2.44) | -3.9 (2.09) |
  Week 36 Change from Baseline: number analyzed (Participants) | 6 | 16 | 11 | 14 | 0
  Week 36 Change from Baseline | -4.2 (1.47) | -3.9 (2.25) | -4.8 (2.09) | -3.9 (2.07) |
  Week 44 Change from Baseline: number analyzed (Participants) | 5 | 15 | 11 | 14 | 0
  Week 44 Change from Baseline | -4.8 (2.39) | -3.7 (2.41) | -4.4 (3.20) | -4.4 (1.95) |
  Week 52 Change from Baseline: number analyzed (Participants) | 4 | 14 | 10 | 14 | 0
  Week 52 Change from Baseline | -3.3 (1.71) | -3.1 (2.40) | -4.2 (2.66) | -4.7 (2.27) |
Statistical Analysis 1: Comparison: APT-1011 1.5 mg HS vs Placebo BID; Least-squares Mean differences, 90% confidence intervals and 1-sided p-values for comparison of each APT-1011 dose group to placebo at Week 12 are from an ANCOVA model; Test type: Other; p = 0.067, ANCOVA; Mean Difference (Final Values) = -1.19, 90% CI 2-sided [-2.49 to 0.12]
Statistical Analysis 2: Comparison: APT-1011 1.5 mg BID vs Placebo BID; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.672, ANCOVA; Mean Difference (Final Values) = 0.34, 90% CI 2-sided [-0.91 to 1.59]
Statistical Analysis 3: Comparison: APT-1011 3 mg HS vs Placebo BID; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.048, ANCOVA; Mean Difference (Final Values) = -1.28, 90% CI 2-sided [-2.55 to -0.01]
Statistical Analysis 4: Comparison: APT-1011 3 mg BID vs Placebo BID; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.653, ANCOVA; Mean Difference (Final Values) = 0.31, 90% CI 2-sided [-0.98 to 1.59]

6. Secondary Outcome: Change in the Number of Dysphagia Episodes
Description: Change in the number of dysphagia episodes at baseline (14-day period prior to randomization) compared with the 14-day period prior to the time point of interest.
  Population used are those who entered Part 1 - Induction. The number of participants analyzed for each timepoint reflect the actual number of participants with data at that timepoint. Note: Following Week 14, all patients in the placebo group were given APT-1011 3mg BID and results reflect the change in the number of dysphagia episodes following 12 or 38 weeks of treatment.
Time Frame: Week 12, Week 26 and Week 52
Population: Full Analysis Set Population receiving double-blind study medication
Measure: Mean (Standard Deviation); unit: change in episodes per 14-day period
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Placebo BID
Number analyzed (Participants) | 18 | 21 | 20 | 19 | 17
change in episodes per 14-day period
  Week 12 Change from Baseline | -8.2 (5.48) | -4.4 (9.41) | -9.3 (7.37) | -9.1 (11.01) | -5.5 (7.89)
  Week 26 Change from Baseline: number analyzed (Participants) | 8 | 19 | 13 | 15 | 0
  Week 26 Change from Baseline | -12.8 (5.65) | -10.0 (10.97) | -9.8 (7.82) | -13.4 (11.78) |
  Week 52 Change from Baseline: number analyzed (Participants) | 5 | 16 | 10 | 14 | 0
  Week 52 Change from Baseline | -11.2 (5.26) | -13.0 (10.79) | -9.5 (9.66) | -14.5 (11.68) |

7. Secondary Outcome: Change From Baseline 7-Day Eosinophilic Esophagitis Activity Index (EEsAI) Total Score
Description: Change from Baseline 7-Day EEsAI total score assessed prior to randomization and those assessed at Weeks 12, 26 and 52 (Total score 100).
  Eosinophilic Esophagitis Activity Index Total Score: 0 (best) to 100 (worst) based on the sum of the categorized subscores for frequency of trouble swallowing [never (0), 1-3x (15) or 4-6x (27) per week]; duration of trouble swallowing [≤5 min (0), >5 min (6)]; pain when swallowing [no (0), yes (15)]; Visual Dysphagia Question score [0 (best),12,19, 21, or 23 (worst)]; avoidance modification and slow eating score [0 (best), 9, or 25 (worst)].
  A higher score means a worse outcome.
  Population used are those who entered Part 1 - Induction. The number of participants analyzed for each timepoint reflect the actual number of participants with data at that timepoint. Note: Following Week 14, all patients in the placebo group were given APT-1011 3mg BID and results reflect the change from baseline 7-day EEs
Time Frame: Weeks 12, 26 and 52
Population: Full Analysis Set Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Placebo BID
Number analyzed (Participants) | 18 | 20 | 20 | 19 | 17
units on a scale
  EEsAI Total Score Week 12 Change from Baseline | -20.4 (15.90) | -15.6 (21.02) | -22.7 (16.60) | -22.6 (21.11) | -9.6 (14.07)
  EEsAI Total Score Week 26 Change from Baseline: number analyzed (Participants) | 8 | 19 | 13 | 16 | 0
  EEsAI Total Score Week 26 Change from Baseline | -25.6 (21.11) | -29.6 (25.48) | -28.8 (21.10) | -34.6 (25.43) |
  EEsAI Total Score Week 52 Change from Baseline: number analyzed (Participants) | 5 | 17 | 11 | 14 | 0
  EEsAI Total Score Week 52 Change from Baseline | -39.8 (28.42) | -37.4 (27.02) | -37.0 (23.72) | -41.1 (20.56) |
Statistical Analysis 1: Comparison: APT-1011 1.5 mg HS vs Placebo BID; EEsAI Total Score Change from Baseline Week 12; Test type: Superiority; p = 0.079, ANCOVA; Mean Difference (Final Values) = -8.81, 90% CI 2-sided [-19.06 to 1.45]
Statistical Analysis 2: Comparison: APT-1011 1.5 mg BID vs Placebo BID; EEsAI Total Score Change from Baseline Week 12; Test type: Superiority; p = 0.195, ANCOVA; Mean Difference (Final Values) = -5.18, 90% CI 2-sided [-15.14 to 4.78]
Statistical Analysis 3: Comparison: APT-1011 3 mg HS vs Placebo BID; EEsAI Total Score Change from Baseline Week 12; Test type: Superiority; p = 0.020, ANCOVA; Mean Difference (Final Values) = -12.56, 90% CI 2-sided [-22.55 to -2.58]
Statistical Analysis 4: Comparison: APT-1011 3 mg BID vs Placebo BID; EEsAI Total Score Change from Baseline Week 12; Test type: Superiority; p = 0.043, ANCOVA; Mean Difference (Final Values) = -10.61, 90% CI 2-sided [-20.74 to -0.48]

8. Secondary Outcome: Change From Baseline 7-Day Eosinophilic Esophagitis Activity Index (EEsAI) Subscores
Description: The Avoidance, Modification and Slow Eating (AMS) Score and Visual Dysphagia Question (VDQ) Score are components of the EEsAI.
  AMS: Answers to three items determining the pattern of behavioral adaptation were scored for each food consistency consumed by the subject (avoidance, modification, and eating slowly). The AMS score ranges from 0 (best) to 25 (worst).
  VDG: The degree of perceived difficulty when eating 8 different food consistencies was assessed. The VDQ score ranges from 0 (best) to 23 (worst).
  A higher score for either subscore means a worse outcome. Negative change from baseline represents a worsening in quality of life for the total score or subscore.
  Population used are those who entered Part 1 - Induction. The number of participants analyzed for each timepoint reflect the actual number of participants with data at that timepoint. Note: Following Week 14, all patients in the placebo group were given APT-1011 3mg BID and results reflect change from baseline.
Time Frame: Weeks 12, 26 and 52
Population: Full Analysis Set Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Placebo BID
Number analyzed (Participants) | 18 | 20 | 20 | 19 | 17
units on a scale
  VDQ Score Week 12 Change from Baseline: number analyzed (Participants) | 18 | 19 | 20 | 19 | 17
  VDQ Score Week 12 Change from Baseline | -3.9 (6.53) | -2.5 (3.24) | -5.0 (6.00) | -4.1 (8.03) | -2.7 (3.41)
  VDQ Score Week 26 Change from Baseline: number analyzed (Participants) | 8 | 18 | 13 | 16 | 0
  VDQ Score Week 26 Change from Baseline | -3.1 (4.36) | -6.8 (7.03) | -6.8 (6.46) | -7.7 (9.47) |
  VDQ Score Week 52 Change from Baseline: number analyzed (Participants) | 5 | 16 | 11 | 14 | 0
  VDQ Score Week 52 Change from Baseline | -9.4 (9.50) | -9.4 (8.25) | -12.6 (9.67) | -9.6 (7.27) |
  AMS Score Week 12 Change from Baseline | 0.0 (0.00) | -3.0 (7.80) | -1.4 (3.30) | -1.3 (6.47) | 1.5 (6.85)
  AMS Score Week 26 Change from Baseline: number analyzed (Participants) | 8 | 19 | 13 | 15 | 0
  AMS Score Week 26 Change from Baseline | 0.0 (0.00) | -2.2 (8.31) | -0.7 (4.44) | -3.3 (7.54) |
  AMS Score Week 52 Change from Baseline: number analyzed (Participants) | 5 | 17 | 11 | 13 | 0
  AMS Score Week 52 Change from Baseline | 0.0 (0.00) | -3.5 (8.39) | -0.8 (2.71) | -2.6 (7.17) |
Statistical Analysis 1: Comparison: APT-1011 1.5 mg HS vs Placebo BID; VDQ Score Change from Baseline Week 12; Test type: Superiority; p = 0.459, ANCOVA; Mean Difference (Final Values) = -0.21, 90% CI 2-sided [-3.49 to 3.08]
Statistical Analysis 2: Comparison: APT-1011 1.5 mg BID vs Placebo BID; VDQ Score Change from Baseline Week 12; Test type: Superiority; p = 0.617, ANCOVA; Mean Difference (Final Values) = 0.58, 90% CI 2-sided [-2.65 to 3.80]
Statistical Analysis 3: Comparison: APT-1011 3 mg HS vs Placebo BID; VDQ Score Change from Baseline Week 12; Test type: Superiority; p = 0.167, ANCOVA; Mean Difference (Final Values) = -1.87, 90% CI 2-sided [-5.07 to 1.33]
Statistical Analysis 4: Comparison: APT-1011 3 mg BID vs Placebo BID; VDQ Score Change from Baseline Week 12; Test type: Superiority; p = 0.373, ANCOVA; Mean Difference (Final Values) = -0.63, 90% CI 2-sided [-3.88 to 2.61]
Statistical Analysis 5: Comparison: APT-1011 1.5 mg HS vs Placebo BID; AMS Score Change from Baseline Week 12; Test type: Superiority; p = 0.203, ANCOVA; Mean Difference (Final Values) = -1.66, 90% CI 2-sided [-4.96 to 1.64]
Statistical Analysis 6: Comparison: APT-1011 1.5 mg BID vs Placebo BID; AMS Score Change from Baseline Week 12; Test type: Superiority; p = 0.014, ANCOVA; Mean Difference (Final Values) = -4.33, 90% CI 2-sided [-7.54 to -1.13]
Statistical Analysis 7: Comparison: APT-1011 3 mg HS vs Placebo BID; AMS Score Change from Baseline Week 12; Test type: Superiority; p = 0.061, ANCOVA; Mean Difference (Final Values) = -3.02, 90% CI 2-sided [-6.23 to 0.20]
Statistical Analysis 8: Comparison: APT-1011 3 mg BID vs Placebo BID; AMS Score Change from Baseline Week 12; Test type: Superiority; p = 0.097, ANCOVA; Mean Difference (Final Values) = -2.57, 90% CI 2-sided [-5.83 to 0.69]

9. Secondary Outcome: Percentage of Subjects With Mean 7-day EEsAI Total Score <20
Description: Percentage of subjects with mean 7-day EEsAI total score <20 to those assessed at Weeks 12, 26 and 52.
  Eosinophilic Esophagitis Activity Index Total Score: 0 (best) to 100 (worst) based on the sum of the categorized subscores for frequency of trouble swallowing [never (0), 1-3x (15) or 4-6x (27) per week]; duration of trouble swallowing [<= 5 min (0), >5 min (6)]; pain when swallowing [no (0), yes (15)]; Visual Dysphagia Question score [0 (best),12,19,21, or 23 (worst)]; avoidance modification and slow eating score [0 (best), 9, or 25 (worst)].
  Population used are those who entered Part 1 - Induction. The number of participants analyzed for each timepoint reflect the actual number of participants with data at that timepoint. Note: Following Week 14, all patients in the placebo group were given APT-1011 3mg BID and results reflect change from baseline global EOE symptom score following 12 or 38 weeks of treatment
Time Frame: Weeks 12, 26, and 52
Population: Full Analysis Set population
Measure: Count of Participants; unit: Participants
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Placebo BID
Number analyzed (Participants) | 18 | 20 | 20 | 19 | 17
Participants
  Week 12 EEsAI Total Score <20 | 4 | 1 | 6 | 5 | 2
  Week 26 EEsAI Total Score <20: number analyzed (Participants) | 8 | 19 | 13 | 16 | 0
  Week 26 EEsAI Total Score <20 | 3 | 5 | 7 | 7 |
  Week 52 EEsAI Total Score <20: number analyzed (Participants) | 5 | 17 | 11 | 14 | 0
  Week 52 EEsAI Total Score <20 | 3 | 7 | 7 | 10 |

10. Secondary Outcome: Change From Baseline Patient Global Impression of Severity (PGIS) for EoE Symptoms as Assessed Prior to Randomization Post-Baseline Visit
Description: Change From Baseline PGIS for EoE Symptoms as Assessed Prior to Randomization at Weeks 4, 8, 12, 14, 18, 22, 26, 28, 36, 44, and 52.
  Population used are those who entered Part 1 - Induction. The number of participants analyzed for each timepoint reflect the actual number of participants with data at that timepoint. Note: Following Week 14, all patients in the placebo group were given APT-1011 3mg BID and results reflect change from baseline global EOE symptoms following 4, 8, 12, 14, 22, 30 or 38 weeks of treatment.
Time Frame: Weeks 4, 8, 12, 14, 18, 22, 26, 28, 36, 44, and 52
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Placebo BID
Number analyzed (Participants) | 20 | 21 | 20 | 19 | 17
Participants
  Week 4: number analyzed (Participants) | 20 | 19 | 20 | 19 | 15
  Week 4: Mild to None | 1 | 0 | 0 | 0 | 1
  Week 4: Mild to Mild | 0 | 0 | 1 | 0 | 0
  Week 4: Mild to Moderate | 0 | 0 | 0 | 0 | 0
  Week 4: Mild to Severe | 1 | 0 | 0 | 0 | 0
  Week 4: Mild to Very Severe | 0 | 0 | 0 | 0 | 0
  Week 4: Moderate to None | 0 | 0 | 4 | 0 | 1
  Week 4: Moderate to Mild | 8 | 7 | 5 | 6 | 5
  Week 4: Moderate to Moderate | 5 | 5 | 4 | 7 | 3
  Week 4: Moderate to Severe | 0 | 0 | 0 | 1 | 0
  Week 4: Moderate to Very Severe | 0 | 0 | 0 | 0 | 0
  Week 4: Severe to None | 0 | 0 | 1 | 0 | 0
  Week 4: Severe to Mild | 3 | 1 | 1 | 1 | 0
  Week 4: Severe to Moderate | 1 | 3 | 3 | 4 | 2
  Week 4: Severe to Severe | 0 | 3 | 1 | 0 | 3
  Week 4: Severe to Very Severe | 0 | 0 | 0 | 0 | 0
  Week 4: Very Severe to None | 0 | 0 | 0 | 0 | 0
  Week 4: Very Severe to Mild | 0 | 0 | 0 | 0 | 0
  Week 4: Very Severe to Moderate | 0 | 0 | 0 | 0 | 0
  Week 4: Very Severe to Severe | 0 | 0 | 0 | 0 | 0
  Week 4: Very Severe to Very Severe | 1 | 0 | 0 | 0 | 0
  Week 8: number analyzed (Participants) | 17 | 21 | 19 | 19 | 16
  Week 8: Mild to None | 0 | 0 | 0 | 0 | 0
  Week 8: Mild to Mild | 0 | 0 | 1 | 0 | 1
  Week 8: Mild to Moderate | 1 | 0 | 0 | 0 | 0
  Week 8: Mild to Severe | 0 | 0 | 0 | 0 | 0
  Week 8: Mild to Very Severe | 0 | 0 | 0 | 0 | 0
  Week 8: Moderate to None | 1 | 1 | 4 | 2 | 1
  Week 8: Moderate to Mild | 8 | 6 | 5 | 6 | 7
  Week 8: Moderate to Moderate | 3 | 6 | 3 | 6 | 2
  Week 8: Moderate to Severe | 0 | 0 | 0 | 0 | 0
  Week 8: Moderate to Very Severe | 0 | 0 | 0 | 0 | 0
  Week 8: Severe to None | 1 | 0 | 1 | 1 | 0
  Week 8: Severe to Mild | 1 | 1 | 2 | 0 | 0
  Week 8: Severe to Moderate | 1 | 6 | 1 | 4 | 5
  Week 8: Severe to Severe | 0 | 1 | 2 | 0 | 0
  Week 8: Severe to Very Severe | 0 | 0 | 0 | 0 | 0
  Week 8: Very Severe to None | 0 | 0 | 0 | 0 | 0
  Week 8: Very Severe to Mild | 0 | 0 | 0 | 0 | 0
  Week 8: Very Severe to Moderate | 0 | 0 | 0 | 0 | 0
  Week 8: Very Severe to Severe | 1 | 0 | 0 | 0 | 0
  Week 8: Very Severe to Very Severe | 0 | 0 | 0 | 0 | 0
  Week 12: number analyzed (Participants) | 18 | 20 | 20 | 18 | 17
  Week 12: Mild to None | 0 | 0 | 0 | 0 | 1
  Week 12: Mild to Mild | 1 | 0 | 1 | 0 | 0
  Week 12: Mild to Moderate | 0 | 0 | 0 | 0 | 0
  Week 12: Mild to Severe | 0 | 0 | 0 | 0 | 0
  Week 12: Mild to Very Severe | 0 | 0 | 0 | 0 | 0
  Week 12: Moderate to None | 1 | 0 | 5 | 2 | 1
  Week 12: Moderate to Mild | 10 | 7 | 5 | 6 | 6
  Week 12: Moderate to Moderate | 2 | 5 | 3 | 4 | 3
  Week 12: Moderate to Severe | 0 | 0 | 0 | 1 | 0
  Week 12: Moderate to Very Severe | 0 | 0 | 0 | 0 | 0
  Week 12: Severe to None | 2 | 0 | 1 | 1 | 0
  Week 12: Severe to Mild | 1 | 3 | 0 | 1 | 1
  Week 12: Severe to Moderate | 0 | 4 | 4 | 2 | 4
  Week 12: Severe to Severe | 0 | 1 | 1 | 1 | 1
  Week 12: Severe to Very Severe | 0 | 0 | 0 | 0 | 0
  Week 12: Very Severe to None | 0 | 0 | 0 | 0 | 0
  Week 12: Very Severe to Mild | 0 | 0 | 0 | 0 | 0
  Week 12: Very Severe to Moderate | 1 | 0 | 0 | 0 | 0
  Week 12: Very Severe to Severe | 0 | 0 | 0 | 0 | 0
  Week 12: Very Severe to Very Severe | 0 | 0 | 0 | 0 | 0
  Week 14: number analyzed (Participants) | 10 | 18 | 13 | 15 | 0
  Week 14: Mild to None | 0 | 0 | 0 | 0 |
  Week 14: Mild to Mild | 1 | 0 | 1 | 0 |
  Week 14: Mild to Moderate | 0 | 0 | 0 | 0 |
  Week 14: Mild to Severe | 0 | 0 | 0 | 0 |
  Week 14: Mild to Very Severe | 0 | 0 | 0 | 0 |
  Week 14: Moderate to None | 0 | 1 | 5 | 4 |
  Week 14: Moderate to Mild | 7 | 8 | 1 | 3 |
  Week 14: Moderate to Moderate | 0 | 2 | 1 | 4 |
  Week 14: Moderate to Severe | 0 | 0 | 0 | 0 |
  Week 14: Moderate to Very Severe | 0 | 0 | 0 | 0 |
  Week 14: Severe to None | 0 | 1 | 0 | 1 |
  Week 14: Severe to Mild | 1 | 1 | 3 | 1 |
  Week 14: Severe to Moderate | 0 | 5 | 1 | 2 |
  Week 14: Severe to Severe | 0 | 0 | 1 | 0 |
  Week 14: Severe to Very Severe | 0 | 0 | 0 | 0 |
  Week 14: Very Severe to None | 0 | 0 | 0 | 0 |
  Week 14: Very Severe to Mild | 0 | 0 | 0 | 0 |
  Week 14: Very Severe to Moderate | 0 | 0 | 0 | 0 |
  Week 14: Very Severe to Severe | 0 | 0 | 0 | 0 |
  Week 14: Very Severe to Very Severe | 1 | 0 | 0 | 0 |
  Week 18: number analyzed (Participants) | 9 | 18 | 14 | 14 | 0
  Week 18: Mild to None | 0 | 0 | 0 | 0 |
  Week 18: Mild to Mild | 0 | 0 | 1 | 0 |
  Week 18: Mild to Moderate | 0 | 0 | 0 | 0 |
  Week 18: Mild to Severe | 0 | 0 | 0 | 0 |
  Week 18: Mild to Very Severe | 0 | 0 | 0 | 0 |
  Week 18: Moderate to None | 0 | 1 | 5 | 5 |
  Week 18: Moderate to Mild | 6 | 9 | 2 | 4 |
  Week 18: Moderate to Moderate | 1 | 1 | 1 | 2 |
  Week 18: Moderate to Severe | 0 | 0 | 0 | 0 |
  Week 18: Moderate to Very Severe | 0 | 0 | 0 | 0 |
  Week 18: Severe to None | 0 | 2 | 1 | 0 |
  Week 18: Severe to Mild | 1 | 2 | 2 | 1 |
  Week 18: Severe to Moderate | 0 | 3 | 1 | 2 |
  Week 18: Severe to Severe | 0 | 0 | 1 | 0 |
  Week 18: Severe to Very Severe | 0 | 0 | 0 | 0 |
  Week 18: Very Severe to None | 0 | 0 | 0 | 0 |
  Week 18: Very Severe to Mild | 0 | 0 | 0 | 0 |
  Week 18: Very Severe to Moderate | 1 | 0 | 0 | 0 |
  Week 18: Very Severe to Severe | 0 | 0 | 0 | 0 |
  Week 18: Very Severe to Very Severe | 0 | 0 | 0 | 0 |
  Week 22: number analyzed (Participants) | 8 | 18 | 13 | 16 | 0
  Week 22: Mild to None | 0 | 0 | 0 | 0 |
  Week 22: Mild to Mild | 0 | 0 | 1 | 0 |
  Week 22: Mild to Moderate | 0 | 0 | 0 | 0 |
  Week 22: Mild to Severe | 0 | 0 | 0 | 0 |
  Week 22: Mild to Very Severe | 0 | 0 | 0 | 0 |
  Week 22: Moderate to None | 1 | 2 | 3 | 4 |
  Week 22: Moderate to Mild | 6 | 8 | 2 | 3 |
  Week 22: Moderate to Moderate | 0 | 1 | 2 | 5 |
  Week 22: Moderate to Severe | 0 | 0 | 0 | 0 |
  Week 22: Moderate to Very Severe | 0 | 0 | 0 | 0 |
  Week 22: Severe to None | 0 | 1 | 1 | 2 |
  Week 22: Severe to Mild | 1 | 3 | 1 | 0 |
  Week 22: Severe to Moderate | 0 | 2 | 2 | 2 |
  Week 22: Severe to Severe | 0 | 1 | 0 | 0 |
  Week 22: Severe to Very Severe | 0 | 0 | 1 | 0 |
  Week 22: Very Severe to None | 0 | 0 | 0 | 0 |
  Week 22: Very Severe to Mild | 0 | 0 | 0 | 0 |
  Week 22: Very Severe to Moderate | 0 | 0 | 0 | 0 |
  Week 22: Very Severe to Severe | 0 | 0 | 0 | 0 |
  Week 22: Very Severe to Very Severe | 0 | 0 | 0 | 0 |
  Week 26: number analyzed (Participants) | 8 | 17 | 13 | 16 | 0
  Week 26: Mild to None | 0 | 0 | 0 | 0 |
  Week 26: Mild to Mild | 0 | 0 | 1 | 0 |
  Week 26: Mild to Moderate | 0 | 0 | 0 | 0 |
  Week 26: Mild to Severe | 0 | 0 | 0 | 0 |
  Week 26: Mild to Very Severe | 0 | 0 | 0 | 0 |
  Week 26: Moderate to None | 2 | 1 | 4 | 5 |
  Week 26: Moderate to Mild | 2 | 8 | 2 | 5 |
  Week 26: Moderate to Moderate | 2 | 2 | 1 | 2 |
  Week 26: Moderate to Severe | 0 | 0 | 0 | 0 |
  Week 26: Moderate to Very Severe | 0 | 0 | 0 | 0 |
  Week 26: Severe to None | 0 | 2 | 2 | 1 |
  Week 26: Severe to Mild | 1 | 2 | 2 | 2 |
  Week 26: Severe to Moderate | 0 | 2 | 0 | 1 |
  Week 26: Severe to Severe | 0 | 0 | 1 | 0 |
  Week 26: Severe to Very Severe | 0 | 0 | 0 | 0 |
  Week 26: Very Severe to None | 0 | 0 | 0 | 0 |
  Week 26: Very Severe to Mild | 0 | 0 | 0 | 0 |
  Week 26: Very Severe to Moderate | 1 | 0 | 0 | 0 |
  Week 26: Very Severe to Severe | 0 | 0 | 0 | 0 |
  Week 26: Very Severe to Very Severe | 0 | 0 | 0 | 0 |
  Week 28: number analyzed (Participants) | 7 | 16 | 10 | 14 | 0
  Week 28: Mild to None | 0 | 0 | 0 | 0 |
  Week 28: Mild to Mild | 0 | 0 | 1 | 0 |
  Week 28: Mild to Moderate | 0 | 0 | 0 | 0 |
  Week 28: Mild to Severe | 0 | 0 | 0 | 0 |
  Week 28: Mild to Very Severe | 0 | 0 | 0 | 0 |
  Week 28: Moderate to None | 2 | 1 | 4 | 4 |
  Week 28: Moderate to Mild | 3 | 7 | 1 | 5 |
  Week 28: Moderate to Moderate | 0 | 2 | 0 | 1 |
  Week 28: Moderate to Severe | 0 | 0 | 0 | 0 |
  Week 28: Moderate to Very Severe | 0 | 0 | 0 | 0 |
  Week 28: Severe to None | 0 | 2 | 2 | 1 |
  Week 28: Severe to Mild | 1 | 2 | 0 | 3 |
  Week 28: Severe to Moderate | 0 | 2 | 1 | 0 |
  Week 28: Severe to Severe | 0 | 0 | 1 | 0 |
  Week 28: Severe to Very Severe | 0 | 0 | 0 | 0 |
  Week 28: Very Severe to None | 0 | 0 | 0 | 0 |
  Week 28: Very Severe to Mild | 1 | 0 | 0 | 0 |
  Week 28: Very Severe to Moderate | 0 | 0 | 0 | 0 |
  Week 28: Very Severe to Severe | 0 | 0 | 0 | 0 |
  Week 28: Very Severe to Very Severe | 0 | 0 | 0 | 0 |
  Week 36: number analyzed (Participants) | 6 | 15 | 11 | 14 | 0
  Week 36: Mild to None | 0 | 0 | 0 | 0 |
  Week 36: Mild to Mild | 0 | 0 | 1 | 0 |
  Week 36: Mild to Moderate | 0 | 0 | 0 | 0 |
  Week 36: Mild to Severe | 0 | 0 | 0 | 0 |
  Week 36: Mild to Very Severe | 0 | 0 | 0 | 0 |
  Week 36: Moderate to None | 0 | 2 | 5 | 4 |
  Week 36: Moderate to Mild | 4 | 7 | 1 | 5 |
  Week 36: Moderate to Moderate | 0 | 1 | 0 | 1 |
  Week 36: Moderate to Severe | 0 | 0 | 0 | 0 |
  Week 36: Moderate to Very Severe | 0 | 0 | 0 | 0 |
  Week 36: Severe to None | 0 | 3 | 2 | 1 |
  Week 36: Severe to Mild | 1 | 2 | 1 | 2 |
  Week 36: Severe to Moderate | 0 | 0 | 0 | 1 |
  Week 36: Severe to Severe | 0 | 0 | 0 | 0 |
  Week 36: Severe to Very Severe | 0 | 0 | 1 | 0 |
  Week 36: Very Severe to None | 0 | 0 | 0 | 0 |
  Week 36: Very Severe to Mild | 0 | 0 | 0 | 0 |
  Week 36: Very Severe to Moderate | 1 | 0 | 0 | 0 |
  Week 36: Very Severe to Severe | 0 | 0 | 0 | 0 |
  Week 36: Very Severe to Very Severe | 0 | 0 | 0 | 0 |
  Week 44: number analyzed (Participants) | 5 | 15 | 10 | 14 | 0
  Week 44: Mild to None | 0 | 0 | 0 | 0 |
  Week 44: Mild to Mild | 0 | 0 | 1 | 0 |
  Week 44: Mild to Moderate | 0 | 0 | 0 | 0 |
  Week 44: Mild to Severe | 0 | 0 | 0 | 0 |
  Week 44: Mild to Very Severe | 0 | 0 | 0 | 0 |
  Week 44: Moderate to None | 1 | 1 | 3 | 5 |
  Week 44: Moderate to Mild | 2 | 8 | 1 | 4 |
  Week 44: Moderate to Moderate | 0 | 1 | 1 | 1 |
  Week 44: Moderate to Severe | 0 | 0 | 0 | 0 |
  Week 44: Moderate to Very Severe | 0 | 0 | 0 | 0 |
  Week 44: Severe to None | 0 | 3 | 2 | 2 |
  Week 44: Severe to Mild | 1 | 2 | 1 | 1 |
  Week 44: Severe to Moderate | 0 | 0 | 0 | 1 |
  Week 44: Severe to Severe | 0 | 0 | 0 | 0 |
  Week 44: Severe to Very Severe | 0 | 0 | 1 | 0 |
  Week 44: Very Severe to None | 0 | 0 | 0 | 0 |
  Week 44: Very Severe to Mild | 1 | 0 | 0 | 0 |
  Week 44: Very Severe to Moderate | 0 | 0 | 0 | 0 |
  Week 44: Very Severe to Severe | 0 | 0 | 0 | 0 |
  Week 44: Very Severe to Very Severe | 0 | 0 | 0 | 0 |
  Week 52: number analyzed (Participants) | 4 | 14 | 10 | 14 | 0
  Week 52: Mild to None | 0 | 0 | 1 | 0 |
  Week 52: Mild to Mild | 0 | 0 | 0 | 0 |
  Week 52: Mild to Moderate | 0 | 0 | 0 | 0 |
  Week 52: Mild to Severe | 0 | 0 | 0 | 0 |
  Week 52: Mild to Very Severe | 0 | 0 | 0 | 0 |
  Week 52: Moderate to None | 0 | 3 | 5 | 8 |
  Week 52: Moderate to Mild | 3 | 3 | 1 | 1 |
  Week 52: Moderate to Moderate | 0 | 4 | 0 | 1 |
  Week 52: Moderate to Severe | 0 | 0 | 0 | 0 |
  Week 52: Moderate to Very Severe | 0 | 0 | 0 | 0 |
  Week 52: Severe to None | 0 | 3 | 1 | 3 |
  Week 52: Severe to Mild | 0 | 1 | 1 | 0 |
  Week 52: Severe to Moderate | 1 | 0 | 0 | 1 |
  Week 52: Severe to Severe | 0 | 0 | 0 | 0 |
  Week 52: Severe to Very Severe | 0 | 0 | 1 | 0 |
  Week 52: Very Severe to None | 0 | 0 | 0 | 0 |
  Week 52: Very Severe to Mild | 0 | 0 | 0 | 0 |
  Week 52: Very Severe to Moderate | 0 | 0 | 0 | 0 |
  Week 52: Very Severe to Severe | 0 | 0 | 0 | 0 |
  Week 52: Very Severe to Very Severe | 0 | 0 | 0 | 0 |

11. Secondary Outcome: Change From Baseline PGIS for Difficulty With Food or Pills Going Down as Assessed Prior to Randomization Post-Baseline Visit
Description: Change From Baseline PGIS for Difficulty with Food or Pills Going Down as Assessed Prior to Randomization at Weeks 4, 8, 12, 14, 18, 22, 26, 28, 36, 44, and 52.
  Population used are those who entered Part 1 - Induction. The number of participants analyzed for each timepoint reflect the actual number of participants with data at that timepoint. Note: Following Week 14, all patients in the placebo group were given APT-1011 3mg BID and results reflect change from baseline PGIS for difficulty with food or pills going down following 4, 8, 12, 14, 22, 30 or 38 weeks of treatment.
Time Frame: Weeks 4, 8, 12, 14, 18, 22, 26, 28, 36, 44, and 52
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Placebo BID
Number analyzed (Participants) | 20 | 21 | 20 | 19 | 17
Participants
  Week 4: number analyzed (Participants) | 20 | 19 | 20 | 19 | 15
  Week 4: Mild to None | 2 | 0 | 0 | 0 | 1
  Week 4: Mild to Mild | 1 | 1 | 1 | 1 | 1
  Week 4: Mild to Moderate | 0 | 0 | 1 | 1 | 0
  Week 4: Mild to Severe | 0 | 0 | 0 | 0 | 0
  Week 4: Mild to Very Severe | 0 | 0 | 0 | 0 | 0
  Week 4: Moderate to None | 0 | 0 | 6 | 0 | 0
  Week 4: Moderate to Mild | 6 | 6 | 4 | 7 | 5
  Week 4: Moderate to Moderate | 5 | 4 | 4 | 4 | 4
  Week 4: Moderate to Severe | 1 | 1 | 0 | 0 | 0
  Week 4: Moderate to Very Severe | 0 | 0 | 0 | 0 | 0
  Week 4: Severe to None | 0 | 0 | 1 | 1 | 0
  Week 4: Severe to Mild | 1 | 1 | 0 | 0 | 0
  Week 4: Severe to Moderate | 2 | 2 | 2 | 4 | 1
  Week 4: Severe to Severe | 1 | 4 | 0 | 1 | 3
  Week 4: Severe to Very Severe | 0 | 0 | 1 | 0 | 0
  Week 4: Very Severe to None | 0 | 0 | 0 | 0 | 0
  Week 4: Very Severe to Mild | 0 | 0 | 0 | 0 | 0
  Week 4: Very Severe to Moderate | 0 | 0 | 0 | 0 | 0
  Week 4: Very Severe to Severe | 0 | 0 | 0 | 0 | 0
  Week 4: Very Severe to Very Severe | 1 | 0 | 0 | 0 | 0
  Week 8: number analyzed (Participants) | 17 | 21 | 19 | 19 | 16
  Week 8: Mild to None | 0 | 0 | 0 | 0 | 1
  Week 8: Mild to Mild | 2 | 1 | 2 | 1 | 2
  Week 8: Mild to Moderate | 1 | 0 | 0 | 1 | 0
  Week 8: Mild to Severe | 0 | 0 | 0 | 0 | 0
  Week 8: Mild to Very Severe | 0 | 0 | 0 | 0 | 0
  Week 8: Moderate to None | 1 | 1 | 4 | 2 | 0
  Week 8: Moderate to Mild | 8 | 5 | 5 | 5 | 6
  Week 8: Moderate to Moderate | 1 | 6 | 4 | 4 | 3
  Week 8: Moderate to Severe | 0 | 0 | 0 | 0 | 0
  Week 8: Moderate to Very Severe | 0 | 0 | 0 | 0 | 0
  Week 8: Severe to None | 1 | 0 | 1 | 1 | 0
  Week 8: Severe to Mild | 2 | 1 | 1 | 2 | 1
  Week 8: Severe to Moderate | 0 | 7 | 0 | 3 | 3
  Week 8: Severe to Severe | 0 | 0 | 1 | 0 | 0
  Week 8: Severe to Very Severe | 0 | 0 | 1 | 0 | 0
  Week 8: Very Severe to None | 0 | 0 | 0 | 0 | 0
  Week 8: Very Severe to Mild | 0 | 0 | 0 | 0 | 0
  Week 8: Very Severe to Moderate | 1 | 0 | 0 | 0 | 0
  Week 8: Very Severe to Severe | 0 | 0 | 0 | 0 | 0
  Week 8: Very Severe to Very Severe | 0 | 0 | 0 | 0 | 0
  Week 12: number analyzed (Participants) | 18 | 20 | 20 | 18 | 17
  Week 12: Mild to None | 1 | 0 | 0 | 0 | 2
  Week 12: Mild to Mild | 2 | 1 | 2 | 2 | 1
  Week 12: Mild to Moderate | 1 | 0 | 0 | 0 | 0
  Week 12: Mild to Severe | 0 | 0 | 0 | 0 | 0
  Week 12: Mild to Very Severe | 0 | 0 | 0 | 0 | 0
  Week 12: Moderate to None | 3 | 0 | 5 | 3 | 0
  Week 12: Moderate to Mild | 4 | 5 | 6 | 2 | 6
  Week 12: Moderate to Moderate | 3 | 6 | 3 | 5 | 4
  Week 12: Moderate to Severe | 0 | 0 | 0 | 0 | 0
  Week 12: Moderate to Very Severe | 0 | 0 | 0 | 0 | 0
  Week 12: Severe to None | 3 | 0 | 1 | 1 | 0
  Week 12: Severe to Mild | 0 | 4 | 0 | 1 | 1
  Week 12: Severe to Moderate | 0 | 3 | 2 | 2 | 2
  Week 12: Severe to Severe | 0 | 1 | 1 | 2 | 1
  Week 12: Severe to Very Severe | 0 | 0 | 0 | 0 | 0
  Week 12: Very Severe to None | 0 | 0 | 0 | 0 | 0
  Week 12: Very Severe to Mild | 0 | 0 | 0 | 0 | 0
  Week 12: Very Severe to Moderate | 1 | 0 | 0 | 0 | 0
  Week 12: Very Severe to Severe | 0 | 0 | 0 | 0 | 0
  Week 12: Very Severe to Very Severe | 0 | 0 | 0 | 0 | 0
  Week 14: number analyzed (Participants) | 10 | 18 | 13 | 15 | 0
  Week 14: Mild to None | 0 | 0 | 1 | 0 |
  Week 14: Mild to Mild | 1 | 1 | 0 | 2 |
  Week 14: Mild to Moderate | 0 | 0 | 0 | 0 |
  Week 14: Mild to Severe | 0 | 0 | 0 | 0 |
  Week 14: Mild to Very Severe | 0 | 0 | 0 | 0 |
  Week 14: Moderate to None | 1 | 0 | 4 | 3 |
  Week 14: Moderate to Mild | 7 | 7 | 3 | 2 |
  Week 14: Moderate to Moderate | 0 | 2 | 1 | 3 |
  Week 14: Moderate to Severe | 0 | 1 | 0 | 0 |
  Week 14: Moderate to Very Severe | 0 | 0 | 0 | 0 |
  Week 14: Severe to None | 0 | 1 | 0 | 1 |
  Week 14: Severe to Mild | 0 | 2 | 2 | 2 |
  Week 14: Severe to Moderate | 0 | 4 | 1 | 2 |
  Week 14: Severe to Severe | 0 | 0 | 1 | 0 |
  Week 14: Severe to Very Severe | 0 | 0 | 0 | 0 |
  Week 14: Very Severe to None | 0 | 0 | 0 | 0 |
  Week 14: Very Severe to Mild | 0 | 0 | 0 | 0 |
  Week 14: Very Severe to Moderate | 0 | 0 | 0 | 0 |
  Week 14: Very Severe to Severe | 0 | 0 | 0 | 0 |
  Week 14: Very Severe to Very Severe | 1 | 0 | 0 | 0 |
  Week 18: number analyzed (Participants) | 9 | 18 | 14 | 14 | 0
  Week 18: Mild to None | 0 | 0 | 1 | 0 |
  Week 18: Mild to Mild | 0 | 1 | 0 | 2 |
  Week 18: Mild to Moderate | 0 | 0 | 0 | 0 |
  Week 18: Mild to Severe | 0 | 0 | 0 | 0 |
  Week 18: Mild to Very Severe | 0 | 0 | 0 | 0 |
  Week 18: Moderate to None | 0 | 1 | 5 | 4 |
  Week 18: Moderate to Mild | 8 | 7 | 3 | 2 |
  Week 18: Moderate to Moderate | 0 | 2 | 1 | 2 |
  Week 18: Moderate to Severe | 0 | 0 | 0 | 0 |
  Week 18: Moderate to Very Severe | 0 | 0 | 0 | 0 |
  Week 18: Severe to None | 0 | 2 | 1 | 1 |
  Week 18: Severe to Mild | 0 | 2 | 1 | 2 |
  Week 18: Severe to Moderate | 0 | 3 | 1 | 1 |
  Week 18: Severe to Severe | 0 | 0 | 1 | 0 |
  Week 18: Severe to Very Severe | 0 | 0 | 0 | 0 |
  Week 18: Very Severe to None | 0 | 0 | 0 | 0 |
  Week 18: Very Severe to Mild | 0 | 0 | 0 | 0 |
  Week 18: Very Severe to Moderate | 1 | 0 | 0 | 0 |
  Week 18: Very Severe to Severe | 0 | 0 | 0 | 0 |
  Week 18: Very Severe to Very Severe | 0 | 0 | 0 | 0 |
  Week 22: number analyzed (Participants) | 8 | 18 | 13 | 16 | 0
  Week 22: Mild to None | 0 | 0 | 0 | 0 |
  Week 22: Mild to Mild | 0 | 1 | 1 | 2 |
  Week 22: Mild to Moderate | 0 | 0 | 0 | 0 |
  Week 22: Mild to Severe | 0 | 0 | 0 | 0 |
  Week 22: Mild to Very Severe | 0 | 0 | 0 | 0 |
  Week 22: Moderate to None | 2 | 1 | 3 | 4 |
  Week 22: Moderate to Mild | 6 | 7 | 3 | 3 |
  Week 22: Moderate to Moderate | 0 | 2 | 2 | 2 |
  Week 22: Moderate to Severe | 0 | 0 | 0 | 0 |
  Week 22: Moderate to Very Severe | 0 | 0 | 0 | 0 |
  Week 22: Severe to None | 0 | 2 | 1 | 2 |
  Week 22: Severe to Mild | 0 | 2 | 1 | 1 |
  Week 22: Severe to Moderate | 0 | 3 | 1 | 2 |
  Week 22: Severe to Severe | 0 | 0 | 0 | 0 |
  Week 22: Severe to Very Severe | 0 | 0 | 1 | 0 |
  Week 22: Very Severe to None | 0 | 0 | 0 | 0 |
  Week 22: Very Severe to Mild | 0 | 0 | 0 | 0 |
  Week 22: Very Severe to Moderate | 0 | 0 | 0 | 0 |
  Week 22: Very Severe to Severe | 0 | 0 | 0 | 0 |
  Week 22: Very Severe to Very Severe | 0 | 0 | 0 | 0 |
  Week 26: number analyzed (Participants) | 8 | 17 | 13 | 16 | 0
  Week 26: Mild to None | 0 | 0 | 0 | 0 |
  Week 26: Mild to Mild | 0 | 1 | 1 | 2 |
  Week 26: Mild to Moderate | 0 | 0 | 0 | 0 |
  Week 26: Mild to Severe | 0 | 0 | 0 | 0 |
  Week 26: Mild to Very Severe | 0 | 0 | 0 | 0 |
  Week 26: Moderate to None | 3 | 0 | 4 | 5 |
  Week 26: Moderate to Mild | 3 | 7 | 3 | 2 |
  Week 26: Moderate to Moderate | 1 | 2 | 1 | 2 |
  Week 26: Moderate to Severe | 0 | 0 | 0 | 0 |
  Week 26: Moderate to Very Severe | 0 | 0 | 0 | 0 |
  Week 26: Severe to None | 0 | 3 | 2 | 2 |
  Week 26: Severe to Mild | 0 | 3 | 1 | 2 |
  Week 26: Severe to Moderate | 0 | 1 | 0 | 1 |
  Week 26: Severe to Severe | 0 | 0 | 1 | 0 |
  Week 26: Severe to Very Severe | 0 | 0 | 0 | 0 |
  Week 26: Very Severe to None | 0 | 0 | 0 | 0 |
  Week 26: Very Severe to Mild | 0 | 0 | 0 | 0 |
  Week 26: Very Severe to Moderate | 1 | 0 | 0 | 0 |
  Week 26: Very Severe to Severe | 0 | 0 | 0 | 0 |
  Week 26: Very Severe to Very Severe | 0 | 0 | 0 | 0 |
  Week 28: number analyzed (Participants) | 7 | 16 | 10 | 14 | 0
  Week 28: Mild to None | 0 | 0 | 1 | 1 |
  Week 28: Mild to Mild | 0 | 1 | 0 | 1 |
  Week 28: Mild to Moderate | 0 | 0 | 0 | 0 |
  Week 28: Mild to Severe | 0 | 0 | 0 | 0 |
  Week 28: Mild to Very Severe | 0 | 0 | 0 | 0 |
  Week 28: Moderate to None | 4 | 0 | 4 | 4 |
  Week 28: Moderate to Mild | 2 | 7 | 1 | 2 |
  Week 28: Moderate to Moderate | 0 | 1 | 0 | 1 |
  Week 28: Moderate to Severe | 0 | 0 | 0 | 0 |
  Week 28: Moderate to Very Severe | 0 | 0 | 0 | 0 |
  Week 28: Severe to None | 0 | 3 | 2 | 1 |
  Week 28: Severe to Mild | 0 | 2 | 0 | 4 |
  Week 28: Severe to Moderate | 0 | 2 | 1 | 0 |
  Week 28: Severe to Severe | 0 | 0 | 1 | 0 |
  Week 28: Severe to Very Severe | 0 | 0 | 0 | 0 |
  Week 28: Very Severe to None | 0 | 0 | 0 | 0 |
  Week 28: Very Severe to Mild | 1 | 0 | 0 | 0 |
  Week 28: Very Severe to Moderate | 0 | 0 | 0 | 0 |
  Week 28: Very Severe to Severe | 0 | 0 | 0 | 0 |
  Week 28: Very Severe to Very Severe | 0 | 0 | 0 | 0 |
  Week 36: number analyzed (Participants) | 6 | 15 | 11 | 14 | 0
  Week 36: Mild to None | 0 | 0 | 0 | 2 |
  Week 36: Mild to Mild | 0 | 1 | 1 | 0 |
  Week 36: Mild to Moderate | 0 | 0 | 0 | 0 |
  Week 36: Mild to Severe | 0 | 0 | 0 | 0 |
  Week 36: Mild to Very Severe | 0 | 0 | 0 | 0 |
  Week 36: Moderate to None | 2 | 2 | 5 | 4 |
  Week 36: Moderate to Mild | 3 | 5 | 1 | 2 |
  Week 36: Moderate to Moderate | 0 | 1 | 0 | 1 |
  Week 36: Moderate to Severe | 0 | 0 | 0 | 0 |
  Week 36: Moderate to Very Severe | 0 | 0 | 0 | 0 |
  Week 36: Severe to None | 0 | 4 | 2 | 1 |
  Week 36: Severe to Mild | 0 | 1 | 1 | 3 |
  Week 36: Severe to Moderate | 0 | 1 | 0 | 1 |
  Week 36: Severe to Severe | 0 | 0 | 0 | 0 |
  Week 36: Severe to Very Severe | 0 | 0 | 1 | 0 |
  Week 36: Very Severe to None | 0 | 0 | 0 | 0 |
  Week 36: Very Severe to Mild | 0 | 0 | 0 | 0 |
  Week 36: Very Severe to Moderate | 0 | 0 | 0 | 0 |
  Week 36: Very Severe to Severe | 1 | 0 | 0 | 0 |
  Week 36: Very Severe to Very Severe | 0 | 0 | 0 | 0 |
  Week 44: number analyzed (Participants) | 5 | 15 | 10 | 14 | 0
  Week 44: Mild to None | 0 | 0 | 0 | 1 |
  Week 44: Mild to Mild | 0 | 1 | 1 | 1 |
  Week 44: Mild to Moderate | 0 | 0 | 0 | 0 |
  Week 44: Mild to Severe | 0 | 0 | 0 | 0 |
  Week 44: Mild to Very Severe | 0 | 0 | 0 | 0 |
  Week 44: Moderate to None | 2 | 1 | 3 | 4 |
  Week 44: Moderate to Mild | 2 | 6 | 1 | 2 |
  Week 44: Moderate to Moderate | 0 | 0 | 1 | 1 |
  Week 44: Moderate to Severe | 0 | 1 | 0 | 0 |
  Week 44: Moderate to Very Severe | 0 | 0 | 0 | 0 |
  Week 44: Severe to None | 0 | 3 | 2 | 2 |
  Week 44: Severe to Mild | 0 | 3 | 1 | 2 |
  Week 44: Severe to Moderate | 0 | 0 | 0 | 1 |
  Week 44: Severe to Severe | 0 | 0 | 0 | 0 |
  Week 44: Severe to Very Severe | 0 | 0 | 1 | 0 |
  Week 44: Very Severe to None | 0 | 0 | 0 | 0 |
  Week 44: Very Severe to Mild | 1 | 0 | 0 | 0 |
  Week 44: Very Severe to Moderate | 0 | 0 | 0 | 0 |
  Week 44: Very Severe to Severe | 0 | 0 | 0 | 0 |
  Week 44: Very Severe to Very Severe | 0 | 0 | 0 | 0 |
  Week 52: number analyzed (Participants) | 4 | 14 | 10 | 14 | 0
  Week 52: Mild to None | 0 | 0 | 1 | 2 |
  Week 52: Mild to Mild | 0 | 0 | 0 | 0 |
  Week 52: Mild to Moderate | 0 | 1 | 0 | 0 |
  Week 52: Mild to Severe | 0 | 0 | 0 | 0 |
  Week 52: Mild to Very Severe | 0 | 0 | 0 | 0 |
  Week 52: Moderate to None | 2 | 2 | 5 | 6 |
  Week 52: Moderate to Mild | 2 | 4 | 1 | 0 |
  Week 52: Moderate to Moderate | 0 | 3 | 0 | 1 |
  Week 52: Moderate to Severe | 0 | 0 | 0 | 0 |
  Week 52: Moderate to Very Severe | 0 | 0 | 0 | 0 |
  Week 52: Severe to None | 0 | 3 | 1 | 3 |
  Week 52: Severe to Mild | 0 | 1 | 1 | 1 |
  Week 52: Severe to Moderate | 0 | 0 | 0 | 1 |
  Week 52: Severe to Severe | 0 | 0 | 0 | 0 |
  Week 52: Severe to Very Severe | 0 | 0 | 1 | 0 |
  Week 52: Very Severe to None | 0 | 0 | 0 | 0 |
  Week 52: Very Severe to Mild | 0 | 0 | 0 | 0 |
  Week 52: Very Severe to Moderate | 0 | 0 | 0 | 0 |
  Week 52: Very Severe to Severe | 0 | 0 | 0 | 0 |
  Week 52: Very Severe to Very Severe | 0 | 0 | 0 | 0 |

12. Secondary Outcome: Change From Baseline Patient Global Impression of Change (PGIC) for EoE Symptoms as Assessed Prior to Randomization Post-Baseline Visit
Description: Change From Baseline PGIC for EoE Symptoms as Assessed Prior to Randomization at Weeks 4, 8, 12, 14, 18, 22, 26, 28, 36, 44, and 52.
  Population used are those who entered Part 1 - Induction. The number of participants analyzed for each timepoint reflect the actual number of participants with data at that timepoint. Note: Following Week 14, all patients in the placebo group were given APT-1011 3mg BID and results reflect change from baseline PGIC for EoE symptoms following 4, 8, 12, 14, 22, 30 or 38 weeks of treatment.
Time Frame: Weeks 4, 8, 12, 14, 18, 22, 26, 36, 44, and 52
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Placebo BID
Number analyzed (Participants) | 21 | 22 | 20 | 20 | 17
Participants
  Week 4: number analyzed (Participants) | 21 | 20 | 20 | 20 | 16
  Week 4: Much Worse | 0 | 0 | 0 | 0 | 0
  Week 4: Moderately Worse | 0 | 0 | 0 | 0 | 1
  Week 4: A Little Worse | 1 | 0 | 1 | 2 | 0
  Week 4: Stayed the Same | 4 | 4 | 4 | 3 | 6
  Week 4: A Little Improved | 9 | 9 | 4 | 10 | 4
  Week 4: Moderately Improved | 4 | 3 | 6 | 2 | 4
  Week 4: Much Improved | 3 | 4 | 5 | 3 | 1
  Week 8: number analyzed (Participants) | 17 | 22 | 19 | 20 | 16
  Week 8: Much Worse | 0 | 0 | 0 | 0 | 0
  Week 8: Moderately Worse | 0 | 0 | 0 | 0 | 0
  Week 8: A Little Worse | 1 | 0 | 1 | 0 | 0
  Week 8: Stayed the Same | 2 | 3 | 3 | 3 | 3
  Week 8: A Little Improved | 4 | 9 | 5 | 7 | 6
  Week 8: Moderately Improved | 7 | 4 | 4 | 6 | 5
  Week 8: Much Improved | 3 | 6 | 6 | 4 | 2
  Week 12: number analyzed (Participants) | 18 | 22 | 20 | 19 | 17
  Week 12: Much Worse | 0 | 0 | 0 | 0 | 0
  Week 12: Moderately Worse | 0 | 0 | 0 | 1 | 0
  Week 12: A Little Worse | 0 | 0 | 1 | 1 | 1
  Week 12: Stayed the Same | 1 | 4 | 4 | 3 | 4
  Week 12: A Little Improved | 6 | 5 | 2 | 6 | 2
  Week 12: Moderately Improved | 5 | 5 | 4 | 3 | 8
  Week 12: Much Improved | 6 | 8 | 9 | 5 | 2
  Week 14: number analyzed (Participants) | 10 | 18 | 13 | 15 | 0
  Week 14: Much Worse | 0 | 0 | 0 | 0 |
  Week 14: Moderately Worse | 0 | 0 | 0 | 0 |
  Week 14: A Little Worse | 0 | 0 | 1 | 1 |
  Week 14: Stayed the Same | 0 | 3 | 1 | 1 |
  Week 14: A Little Improved | 3 | 4 | 1 | 5 |
  Week 14: Moderately Improved | 5 | 3 | 3 | 3 |
  Week 14: Much Improved | 2 | 8 | 7 | 5 |
  Week 18: number analyzed (Participants) | 9 | 18 | 14 | 14 | 0
  Week 18: Much Worse | 0 | 0 | 0 | 0 |
  Week 18: Moderately Worse | 0 | 0 | 1 | 0 |
  Week 18: A Little Worse | 0 | 1 | 1 | 0 |
  Week 18: Stayed the Same | 0 | 3 | 0 | 1 |
  Week 18: A Little Improved | 2 | 1 | 1 | 4 |
  Week 18: Moderately Improved | 6 | 2 | 1 | 3 |
  Week 18: Much Improved | 1 | 11 | 10 | 6 |
  Week 22: number analyzed (Participants) | 8 | 18 | 14 | 16 | 0
  Week 22: Much Worse | 0 | 0 | 1 | 0 |
  Week 22: Moderately Worse | 0 | 0 | 1 | 0 |
  Week 22: A Little Worse | 0 | 0 | 0 | 1 |
  Week 22: Stayed the Same | 0 | 3 | 0 | 1 |
  Week 22: A Little Improved | 2 | 1 | 2 | 5 |
  Week 22: Moderately Improved | 2 | 3 | 3 | 1 |
  Week 22: Much Improved | 4 | 11 | 7 | 8 |
  Week 26: number analyzed (Participants) | 8 | 18 | 13 | 16 | 0
  Week 26: Much Worse | 0 | 0 | 0 | 0 |
  Week 26: Moderately Worse | 0 | 0 | 2 | 1 |
  Week 26: A Little Worse | 0 | 0 | 0 | 0 |
  Week 26: Stayed the Same | 0 | 2 | 0 | 1 |
  Week 26: A Little Improved | 3 | 1 | 0 | 4 |
  Week 26: Moderately Improved | 1 | 2 | 2 | 0 |
  Week 26: Much Improved | 4 | 13 | 9 | 10 |
  Week 28: number analyzed (Participants) | 7 | 17 | 10 | 14 | 0
  Week 28: Much Worse | 0 | 0 | 0 | 0 |
  Week 28: Moderately Worse | 0 | 0 | 1 | 0 |
  Week 28: A Little Worse | 0 | 0 | 0 | 0 |
  Week 28: Stayed the Same | 0 | 3 | 0 | 0 |
  Week 28: A Little Improved | 1 | 0 | 1 | 2 |
  Week 28: Moderately Improved | 2 | 3 | 0 | 2 |
  Week 28: Much Improved | 4 | 11 | 8 | 10 |
  Week 36: number analyzed (Participants) | 6 | 16 | 11 | 14 | 0
  Week 36: Much Worse | 0 | 0 | 0 | 0 |
  Week 36: Moderately Worse | 0 | 0 | 0 | 0 |
  Week 36: A Little Worse | 0 | 0 | 0 | 0 |
  Week 36: Stayed the Same | 1 | 0 | 1 | 0 |
  Week 36: A Little Improved | 1 | 1 | 0 | 3 |
  Week 36: Moderately Improved | 1 | 1 | 0 | 2 |
  Week 36: Much Improved | 3 | 14 | 10 | 9 |
  Week 44: number analyzed (Participants) | 5 | 15 | 11 | 14 | 0
  Week 44: Much Worse | 0 | 0 | 1 | 0 |
  Week 44: Moderately Worse | 0 | 0 | 0 | 0 |
  Week 44: A Little Worse | 0 | 0 | 0 | 0 |
  Week 44: Stayed the Same | 0 | 0 | 0 | 0 |
  Week 44: A Little Improved | 1 | 2 | 0 | 2 |
  Week 44: Moderately Improved | 1 | 1 | 2 | 2 |
  Week 44: Much Improved | 3 | 12 | 8 | 10 |
  Week 52: number analyzed (Participants) | 4 | 14 | 10 | 14 | 0
  Week 52: Much Worse | 0 | 0 | 0 | 0 |
  Week 52: Moderately Worse | 0 | 0 | 0 | 0 |
  Week 52: A Little Worse | 0 | 0 | 1 | 0 |
  Week 52: Stayed the Same | 0 | 1 | 0 | 0 |
  Week 52: A Little Improved | 1 | 0 | 0 | 2 |
  Week 52: Moderately Improved | 2 | 3 | 1 | 1 |
  Week 52: Much Improved | 1 | 10 | 8 | 11 |

13. Secondary Outcome: Change From Baseline PGIC of Difficulty With Food or Pills as Assessed Prior to Randomization Post-Baseline Visit
Description: Change From Baseline PGIC of Difficulty with Food or Pills as Assessed Prior to Randomization at Weeks 4, 8, 12, 14, 18, 22, 26, 28, 36, 44, and 52.
  Population used are those who entered Part 1 - Induction. The number of participants analyzed for each timepoint reflect the actual number of participants with data at that timepoint. Note: Following Week 14, all patients in the placebo group were given APT-1011 3mg BID and results reflect change from baseline PGIC of difficulty with food or pills following 4, 8, 12, 14, 22, 30 or 38 weeks of treatment.
Time Frame: Weeks 4, 8, 12, 14, 18, 22, 26, 36, 44, and 52
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Placebo BID
Number analyzed (Participants) | 21 | 22 | 20 | 20 | 17
Participants
  Week 4: number analyzed (Participants) | 21 | 20 | 20 | 20 | 16
  Week 4: Much Worse | 0 | 0 | 0 | 0 | 0
  Week 4: Moderately Worse | 0 | 0 | 0 | 0 | 0
  Week 4: A Little Worse | 1 | 0 | 2 | 1 | 1
  Week 4: Stayed the Same | 4 | 3 | 4 | 5 | 5
  Week 4: A Little Improved | 8 | 10 | 4 | 9 | 7
  Week 4: Moderately Improved | 6 | 5 | 4 | 2 | 2
  Week 4: Much Improved | 2 | 2 | 6 | 3 | 1
  Week 8: number analyzed (Participants) | 17 | 22 | 19 | 20 | 16
  Week 8: Much Worse | 0 | 0 | 1 | 0 | 0
  Week 8: Moderately Worse | 0 | 0 | 0 | 0 | 0
  Week 8: A Little Worse | 2 | 0 | 1 | 0 | 1
  Week 8: Stayed the Same | 2 | 5 | 1 | 4 | 4
  Week 8: A Little Improved | 3 | 5 | 5 | 5 | 5
  Week 8: Moderately Improved | 6 | 4 | 3 | 7 | 5
  Week 8: Much Improved | 4 | 8 | 8 | 4 | 1
  Week 12: number analyzed (Participants) | 18 | 22 | 20 | 19 | 17
  Week 12: Much Worse | 0 | 0 | 0 | 0 | 0
  Week 12: Moderately Worse | 0 | 0 | 0 | 1 | 0
  Week 12: A Little Worse | 0 | 0 | 2 | 1 | 0
  Week 12: Stayed the Same | 1 | 4 | 2 | 3 | 3
  Week 12: A Little Improved | 5 | 5 | 5 | 5 | 6
  Week 12: Moderately Improved | 6 | 4 | 2 | 3 | 6
  Week 12: Much Improved | 6 | 9 | 9 | 6 | 2
  Week 14: number analyzed (Participants) | 10 | 18 | 13 | 15 | 0
  Week 14: Much Worse | 0 | 0 | 0 | 0 |
  Week 14: Moderately Worse | 0 | 0 | 0 | 0 |
  Week 14: A Little Worse | 0 | 0 | 2 | 0 |
  Week 14: Stayed the Same | 0 | 4 | 0 | 3 |
  Week 14: A Little Improved | 3 | 3 | 1 | 4 |
  Week 14: Moderately Improved | 4 | 3 | 2 | 3 |
  Week 14: Much Improved | 3 | 8 | 8 | 5 |
  Week 18: number analyzed (Participants) | 9 | 18 | 14 | 14 | 0
  Week 18: Much Worse | 0 | 0 | 0 | 0 |
  Week 18: Moderately Worse | 0 | 0 | 1 | 0 |
  Week 18: A Little Worse | 0 | 1 | 1 | 1 |
  Week 18: Stayed the Same | 0 | 3 | 0 | 0 |
  Week 18: A Little Improved | 1 | 1 | 1 | 2 |
  Week 18: Moderately Improved | 6 | 4 | 2 | 4 |
  Week 18: Much Improved | 2 | 9 | 9 | 7 |
  Week 22: number analyzed (Participants) | 8 | 18 | 14 | 16 | 0
  Week 22: Much Worse | 0 | 0 | 1 | 0 |
  Week 22: Moderately Worse | 0 | 0 | 1 | 0 |
  Week 22: A Little Worse | 0 | 0 | 0 | 1 |
  Week 22: Stayed the Same | 0 | 2 | 0 | 1 |
  Week 22: A Little Improved | 2 | 2 | 2 | 5 |
  Week 22: Moderately Improved | 2 | 5 | 3 | 0 |
  Week 22: Much Improved | 4 | 9 | 7 | 9 |
  Week 26: number analyzed (Participants) | 8 | 18 | 13 | 16 | 0
  Week 26: Much Worse | 0 | 0 | 0 | 0 |
  Week 26: Moderately Worse | 0 | 0 | 2 | 1 |
  Week 26: A Little Worse | 0 | 1 | 0 | 0 |
  Week 26: Stayed the Same | 0 | 2 | 0 | 1 |
  Week 26: A Little Improved | 2 | 0 | 0 | 3 |
  Week 26: Moderately Improved | 4 | 3 | 2 | 1 |
  Week 26: Much Improved | 2 | 12 | 9 | 10 |
  Week 28: number analyzed (Participants) | 7 | 17 | 10 | 14 | 0
  Week 28: Much Worse | 0 | 0 | 0 | 0 |
  Week 28: Moderately Worse | 0 | 0 | 1 | 0 |
  Week 28: A Little Worse | 0 | 0 | 0 | 0 |
  Week 28: Stayed the Same | 0 | 2 | 0 | 0 |
  Week 28: A Little Improved | 1 | 1 | 1 | 1 |
  Week 28: Moderately Improved | 2 | 3 | 0 | 4 |
  Week 28: Much Improved | 4 | 11 | 8 | 9 |
  Week 36: number analyzed (Participants) | 6 | 16 | 11 | 14 | 0
  Week 36: Much Worse | 0 | 0 | 0 | 0 |
  Week 36: Moderately Worse | 0 | 0 | 0 | 0 |
  Week 36: A Little Worse | 0 | 0 | 0 | 0 |
  Week 36: Stayed the Same | 0 | 1 | 1 | 0 |
  Week 36: A Little Improved | 1 | 0 | 0 | 2 |
  Week 36: Moderately Improved | 3 | 3 | 0 | 3 |
  Week 36: Much Improved | 2 | 12 | 10 | 9 |
  Week 44: number analyzed (Participants) | 5 | 15 | 11 | 14 | 0
  Week 44: Much Worse | 0 | 0 | 1 | 0 |
  Week 44: Moderately Worse | 0 | 0 | 0 | 0 |
  Week 44: A Little Worse | 0 | 0 | 0 | 0 |
  Week 44: Stayed the Same | 0 | 1 | 0 | 0 |
  Week 44: A Little Improved | 1 | 0 | 0 | 2 |
  Week 44: Moderately Improved | 1 | 1 | 2 | 2 |
  Week 44: Much Improved | 3 | 13 | 8 | 10 |
  Week 52: number analyzed (Participants) | 4 | 14 | 10 | 14 | 0
  Week 52: Much Worse | 0 | 0 | 0 | 0 |
  Week 52: Moderately Worse | 0 | 0 | 0 | 0 |
  Week 52: A Little Worse | 0 | 1 | 1 | 0 |
  Week 52: Stayed the Same | 1 | 0 | 0 | 0 |
  Week 52: A Little Improved | 0 | 0 | 0 | 2 |
  Week 52: Moderately Improved | 1 | 5 | 1 | 3 |
  Week 52: Much Improved | 2 | 8 | 8 | 9 |

14. Secondary Outcome: Percentage of Histologic Non-responders by Dose at Weeks 12, 26, and 52
Description: Percentage of histologic non-responders by dose at Weeks 12, 26, and 52.
  Note: Following Week 14, all patients in the placebo group were given APT-1011 3mg BID and results reflect non-response following 12 or 38 weeks of treatment.
Time Frame: Weeks 12, 26 and 52
Population: Full Analysis Set Population
Measure: Count of Participants; unit: Participants
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Placebo BID
Number analyzed (Participants) | 21 | 22 | 21 | 20 | 19
Participants
  Week 12 | 11 | 2 | 7 | 4 | 19
  Week 26 | 11 | 5 | 7 | 5 | 7
  Week 52 | 16 | 6 | 10 | 8 | 9

15. Secondary Outcome: Percentage of Subjects Requiring Emergency Endoscopic Food Dis-impaction
Description: Percentage of subjects requiring emergency endoscopic food dis-impaction by dose before Week 14, between Week 14 and Week 28, and between Week 28 and Week 52.
  Note: There were no patients in the placebo group after Week 14.
Time Frame: before Week 14, between Week 14 and Week 28, between Week 28 and Week 52
Population: Full Analysis Set Population
Measure: Count of Participants; unit: Participants
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Placebo BID
Number analyzed (Participants) | 21 | 22 | 21 | 20 | 19
Participants
  Before Week 14 | 0 | 0 | 0 | 0 | 0
  Between Week 14 and Week 28 | 0 | 0 | 0 | 0 | 0
  Between Week 28 and Week 52 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Percentage of Subjects Requiring Esophageal Dilation
Description: Percentage of subjects requiring esophageal dilation by dosing group and part of the study.
  Note: There were no patients in the placebo group after Week 14.
Time Frame: baseline to Week 52
Population: Full Analysis Set Population
Measure: Count of Participants; unit: Participants
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Placebo BID
Number analyzed (Participants) | 21 | 22 | 21 | 20 | 19
Participants | 0 | 0 | 0 | 0 | 0

17. Other Pre Specified Outcome: Number of Subjects Discontinuing Due to HPA Axis Suppression
Description: Number of subjects discontinuing due to HPA axis suppression.
  Note: There were no patients in the placebo group after Week 14.
Time Frame: baseline to Week 52
Population: Safety Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Placebo BID
Number analyzed (Participants) | 21 | 23 | 21 | 20 | 19
Participants | 0 | 0 | 0 | 0 | 0

18. Other Pre Specified Outcome: Number of Subjects With Oral and Esophageal Candidiasis
Description: Frequency of oral and esophageal candidiasis.
  Note: There were no patients in the placebo group after Week 14.
Time Frame: baseline to Week 52
Population: Safety Analysis Population
Measure: Count of Participants; unit: Participants
Groups:
- Single-blind APT-1011 3 mg BID: APT-1011 3 mg after breakfast, APT-1011 3 mg HS
  APT-1011: APT-1011 is an orally disintegrating tablet formulation of fluticasone propionate
- Total APT-1011 3 mg BID: The Total APT-1011 3 mg BID group comprises all subjects who received double-blind or single-blind APT-1011 3 mg BID during Part 2
  APT-1011: APT-1011 is an orally disintegrating tablet formulation of fluticasone propionate
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Placebo BID | Single-blind APT-1011 3 mg BID | Total APT-1011 3 mg BID
Number analyzed (Participants) | 21 | 23 | 21 | 20 | 19 | 34 | 51
Participants
  Oesophageal candidiasis | 0 | 2 | 0 | 8 | 0 | 1 | 9
  Oral candidiasis | 0 | 3 | 1 | 3 | 0 | 1 | 4

19. Other Pre Specified Outcome: Number of Subjects With Treatment-Emergent Adverse Events Leading to Study Discontinuation in Part 1
Description: Number of Subjects With Treatment-Emergent Adverse Events (TEAEs) Leading to Study Discontinuation in Part 1.
Time Frame: baseline to Week 12
Population: Safety Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Placebo BID | Total APT-1011 3 mg BID
Number analyzed (Participants) | 21 | 23 | 21 | 20 | 20 | 85
Participants | 0 | 2 | 0 | 1 | 2 | 3

20. Other Pre Specified Outcome: Number of Subjects With Treatment-Emergent Adverse Events Leading to Study Discontinuation in Part 2
Description: Number of Subjects With Treatment-Emergent Adverse Events (TEAEs) Leading to Study Discontinuation in Part 2.
Time Frame: Week 12 to 52
Population: Safety Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Placebo BID | Single-blind APT-1011 3mg BID | Total APT-1011 3 mg BID
Number analyzed (Participants) | 10 | 19 | 14 | 16 | 0 | 34 | 50
Participants | 1 | 0 | 0 | 0 |  | 0 | 0

21. Other Pre Specified Outcome: Percentage of Subjects With Serum Cortisol Level ≤5 μg/dL or Abnormal Adrenocorticotropic Hormone (ACTH) Stimulation Test
Description: Percentage of subjects with serum cortisol level ≤5 μg/dL (≤138 nmol/L) or abnormal adrenocorticotropic hormone (ACTH) stimulation test (serum cortisol <16 μg/dL [≤440 nmol/L] at 60 minutes).
  Population used are those who entered Part 2 - Maintenance. The number of participants analyzed for each timepoint reflect the actual number of participants with data at that timepoint.
Time Frame: Week 12 to 52
Population: Safety Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | APT-1011 1.5 mg HS | APT-1011 1.5 mg BID | APT-1011 3 mg HS | APT-1011 3 mg BID | Placebo BID
Number analyzed (Participants) | 9 | 19 | 14 | 16 | 0
Participants
  Serum cortisol level <=5 ug/dL (<=138 mmol/L) | 4 | 1 | 4 | 6 | 0
  Abnormal ACTH stimulation test result serum cortisol level <16ug/Dl (<=440 nmol/L): number analyzed (Participants) | 9 | 19 | 13 | 16 | 0
  Abnormal ACTH stimulation test result serum cortisol level <16ug/Dl (<=440 nmol/L) | 0 | 2 | 1 | 4 | 0

ADVERSE EVENTS:
Time Frame: to Week 14 (Part 1) to Week 52 (Part 2)
Description: Adverse events were collected and reported from the time of signature on the ICF to the last study visit. All SAEs were collected and reported from the ICF signature to 30 days after the last study procedure or study drug administration.
  One subject randomized to placebo was erroneously dispensed APT-1011 1.5 mg BID therefore this subject is included in the APT-1011 1.5mg BID arm for safety reporting (FAS). This subject is included in the placebo arm for efficacy reporting (ITT).
Groups:
- APT-1011 1.5 mg HS Part 1: Placebo after breakfast, APT-1011 1.5 mg HS
  APT-1011: APT-1011 is an orally disintegrating tablet formulation of fluticasone propionate
  Placebo: Placebo tablets are identical in composition to APT-1011 except they exclude the active ingredient.
- APT-1011 1.5 mg BID Part 1: APT-1011 1.5 mg after breakfast, APT-1011 1.5 mg HS
  APT-1011: APT-1011 is an orally disintegrating tablet formulation of fluticasone propionate
- APT-1011 3 mg HS Part 1: Placebo after breakfast, APT-1011 3 mg HS
  APT-1011: APT-1011 is an orally disintegrating tablet formulation of fluticasone propionate
  Placebo: Placebo tablets are identical in composition to APT-1011 except they exclude the active ingredient.
- APT-1011 3 mg BID Part 1: APT-1011 3 mg after breakfast, APT-1011 3 mg HS
  APT-1011: APT-1011 is an orally disintegrating tablet formulation of fluticasone propionate
- Placebo BID Part 1: Placebo 30 minutes after breakfast and HS
  Placebo: Placebo tablets are identical in composition to APT-1011 except they exclude the active ingredient.
- Double-blind APT-1011 1.5 mg HS Part 2: Placebo after breakfast, APT-1011 1.5 mg HS
  Histologic responders at Week 12 who continued in Part 2 are included in double-blind dosing groups.
  APT-1011: APT-1011 is an orally disintegrating tablet formulation of fluticasone propionate
  Placebo: Placebo tablets are identical in composition to APT-1011 except they exclude the active ingredient.
- Double-blind APT-1011 1.5 mg BID Part 2: APT-1011 1.5 mg after breakfast, APT-1011 1.5 mg HS
  Histologic responders at Week 12 who continued in Part 2 are included in double-blind dosing groups.
  APT-1011: APT-1011 is an orally disintegrating tablet formulation of fluticasone propionate
- Double-blind APT-1011 3 mg HS Part 2: Placebo after breakfast, APT-1011 3 mg HS
  Histologic responders at Week 12 who continued in Part 2 are included in double-blind dosing groups.
  APT-1011: APT-1011 is an orally disintegrating tablet formulation of fluticasone propionate
  Placebo: Placebo tablets are identical in composition to APT-1011 except they exclude the active ingredient.
- Double-blind APT-1011 3 mg BID Part 2: APT-1011 3 mg after breakfast, APT-1011 3 mg HS
  Histologic responders at Week 12 who continued in Part 2 are included in double-blind dosing groups.
  APT-1011: APT-1011 is an orally disintegrating tablet formulation of fluticasone propionate
- Single-blind APT-1011 3mg BID Part 2: APT-1011 3 mg after breakfast, APT-1011 3 mg HS
  Histologic non-responders at Week 12 who continued in Part 2 are included in the single-blind APT-1011 3 mg BID group.
  APT-1011: APT-1011 is an orally disintegrating tablet formulation of fluticasone propionate
- Total APT-1011 3 mg BID Part 2: The Total APT-1011 3 mg BID group comprises all subjects who received double-blind or single-blind APT-1011 3 mg BID during Part 2
  APT-1011: APT-1011 is an orally disintegrating tablet formulation of fluticasone propionate
Arm/Group | APT-1011 1.5 mg HS Part 1 | APT-1011 1.5 mg BID Part 1 | APT-1011 3 mg HS Part 1 | APT-1011 3 mg BID Part 1 | Placebo BID Part 1 | Double-blind APT-1011 1.5 mg HS Part 2 | Double-blind APT-1011 1.5 mg BID Part 2 | Double-blind APT-1011 3 mg HS Part 2 | Double-blind APT-1011 3 mg BID Part 2 | Single-blind APT-1011 3mg BID Part 2 | Total APT-1011 3 mg BID Part 2
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/23 | 0/21 | 0/20 | 0/20 | 0/10 | 0/19 | 0/14 | 0/16 | 0/34 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/23 | 1/21 | 0/20 | 0/20 | 1/10 | 0/19 | 1/14 | 0/16 | 0/34 | 0/50
Other Adverse Events (participants affected / at risk) | 13/21 | 17/23 | 16/21 | 17/20 | 13/20 | 7/10 | 14/19 | 13/14 | 12/16 | 22/34 | 34/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | APT-1011 1.5 mg HS Part 1 (N=21) | APT-1011 1.5 mg BID Part 1 (N=23) | APT-1011 3 mg HS Part 1 (N=21) | APT-1011 3 mg BID Part 1 (N=20) | Placebo BID Part 1 (N=20) | Double-blind APT-1011 1.5 mg HS Part 2 (N=10) | Double-blind APT-1011 1.5 mg BID Part 2 (N=19) | Double-blind APT-1011 3 mg HS Part 2 (N=14) | Double-blind APT-1011 3 mg BID Part 2 (N=16) | Single-blind APT-1011 3mg BID Part 2 (N=34) | Total APT-1011 3 mg BID Part 2 (N=50)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | APT-1011 1.5 mg HS Part 1 (N=21) | APT-1011 1.5 mg BID Part 1 (N=23) | APT-1011 3 mg HS Part 1 (N=21) | APT-1011 3 mg BID Part 1 (N=20) | Placebo BID Part 1 (N=20) | Double-blind APT-1011 1.5 mg HS Part 2 (N=10) | Double-blind APT-1011 1.5 mg BID Part 2 (N=19) | Double-blind APT-1011 3 mg HS Part 2 (N=14) | Double-blind APT-1011 3 mg BID Part 2 (N=16) | Single-blind APT-1011 3mg BID Part 2 (N=34) | Total APT-1011 3 mg BID Part 2 (N=50)
Nasopharyngitis (Infections and infestations) | 3 | 3 | 2 | 0 | 2 | 2 | 1 | 0 | 5 | 4 | 9
Oeseophageal candidiasis (Infections and infestations) | 0 | 2 | 0 | 6 | 0 | 0 | 1 | 0 | 3 | 1 | 4
Oral candidiasis (Infections and infestations) | 0 | 2 | 1 | 2 | 0 | 0 | 2 | 0 | 2 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 2
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Genital infection fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angular cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Faeces pale (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastric mucosa erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oesophageal food impaction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 1 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cortisol decreased (Investigations) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Protein urine present (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
ACTH stimulation test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Electrocardiogram QRS complex prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neutrophil percentage decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 1 | 3 | 2 | 1 | 1 | 2 | 1 | 2 | 3
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal spasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Generalized oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Temperature regulation disorder (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cutaneous calcification (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Epididymal cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Peyronie's disease (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Libido decreased (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Appetite disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypovitaminosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness bilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Adrenal suppression (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Cartilage neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gilbert's syndrome (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-07-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT03191864/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT03191864/SAP_001.pdf